CLINICAL TRIAL: NCT00669409
Title: A PHASE 1/2A, RANDOMIZED, PLACEBO-CONTROLLED, DOUBLE BLIND, DOSE-ESCALATION, MULTICENTER STUDY OF THE SAFETY, TOLERABILITY, EFFICACY AND PHARMACOKINETICS, OF A SINGLE INTRAVENOUS DOSE OF PF-04383119 IN JAPANESE PATIENTS WITH MODERATE TO SEVERE PAIN FROM OSTEOARTHRITIS OF THE KNEE
Brief Title: A Phase 1/2A, Single Dose Study Of PF-04383119 In Japanese Patients With Moderate To Severe Pain From Osteoarthritis Of The Knee
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A4091022
Record Dates: First submitted 2008-04-25; First posted 2008-04-30 (Estimated); Results first posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-01

CONDITIONS: Osteoarthritis, Knee
Keywords: monoclonal antibody
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — tanezumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- 10 mcg/kg (Experimental)
  Interventions: Drug: PF-04383119 (tanezumab)
- 100 mcg/kg (Experimental)
  Interventions: Drug: PF-04383119 (tanezumab)
- 200 mcg/kg (Experimental)
  Interventions: Drug: PF-04383119 (tanezumab)
- 25 mcg/kg (Experimental)
  Interventions: Drug: PF-04383119 (tanezumab)
- 50 mcg/kg (Experimental)
  Interventions: Drug: PF-04383119 (tanezumab)
- Placebo (Placebo Comparator)
  Interventions: Drug: PF-04383119 (tanezumab)

INTERVENTIONS:
Drug: PF-04383119 (tanezumab) — single dose of 10 mcg/kg IV
  Arms: 10 mcg/kg
Drug: PF-04383119 (tanezumab) — single dose of 100 mcg/kg IV
  Arms: 100 mcg/kg
Drug: PF-04383119 (tanezumab) — single dose of 200 mcg/kg IV
  Arms: 200 mcg/kg
Drug: PF-04383119 (tanezumab) — single dose of 25 mcg/kg IV
  Arms: 25 mcg/kg
Drug: PF-04383119 (tanezumab) — single dose of 50 mcg/kg IV
  Arms: 50 mcg/kg
Drug: PF-04383119 (tanezumab) — single dose of Placebo IV
  Arms: Placebo

SUMMARY:
To evaluate the safety and tolerability of single IV doses of PF-04383119 in Japanese patients with moderate to severe pain from OA of the knee (Part I). To evaluate the preliminary analgesic efficacy of PF-04383119 in Japanese patients with moderate to severe pain from OA of the knee in comparison with placebo (Part I and Part II).

ELIGIBILITY:
Inclusion Criteria:

* Japanese Male or female, Age 35-65 (Part 1), Age 35-75 (Part 2)
* Diagnosis of osteoarthritis (OA) of the knee based on American College of Rheumatology criteria
* Knee pain, and radiographic evidence of knee OA (Kellgren-Lawrence x-ray grade ≥2) obtained within 1 year of enrollment
* At least one of the following: age >50, morning stiffness <30 minutes in duration, crepitus, and OA of the knee must involve the index tibiofemoral joint and must have present for at least 6 months
* Patients who meet at least one of the following: unwilling to take non-opiate pain medications, or for whom non-opiate pain medications have failed, or are candidates for or seeking invasive interventions such as intraarticular injections, knee arthroplasty, or total knee surgery
* Pain levels as required by the protocol at Screening and Baseline

Exclusion Criteria:

* Diagnosis or history of RA, any inflammatory arthritis, gout, Paget's disease or any other disease that in the Investigator's opinion would interfere with the assessment of pain and other symptoms of OA
* Patients with regional pain syndromes suggestive of fibromyalgia or regional pain caused by lumbar or cervical compressions with radiculopathy or at risk of developing radiculopathy.
* Diagnosis or history of fibromyalgia
* Planned surgical procedure during the duration of the study

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2008-06-06 (Actual); Primary Completion 2009-12-25 (Actual); Study Completion 2009-12-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (12):
- Japan (12):
  - National Hospital Organization Takasaki General Medical Center, Takasaki, Gunma
  - Fujisawa shounandai Hospital, Fujisawa-shi, Kanagawa
  - Nippon Kokan Clinic, Kawasaki, Kanagawa
  - Medical Corporation Yamamoto Kinenkai Yamamoto Kinen Hospital, Yokohama, Kanagawa
  - Nakamura Hospital, Beppu-shi, Oita Prefecture
  - Tokyo Metropolitan Fuchu Hospital, Fuchū, Tokyo
  - FuruKawabashi Hospital, Minato-ku, Tokyo
  - Research Hospital, the Institute of Medical Science, the University of Tokyo, Minato-ku, Tokyo
  - Kitashinagawa Third Hospital, Shinagawa-ku, Tokyo
  - Oosaki Hospital Tokyo Heart Center, Shinagawa-ku, Tokyo
  - Kanto Medical Center Ntt Ec, Shinagawa-ku, Tokyo
  - International Medical Center of Japan Toyama Hospital, Shinjuku-ku, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Nagashima H, Suzuki M, Araki S, Yamabe T, Muto C; Tanezumab Investigators. Preliminary assessment of the safety and efficacy of tanezumab in Japanese patients with moderate to severe osteoarthritis of the knee: a randomized, double-blind, dose-escalation, placebo-controlled study. Osteoarthritis Cartilage. 2011 Dec;19(12):1405-12. doi: 10.1016/j.joca.2011.09.006. Epub 2011 Oct 5. PMID 22004765

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 83 participants were enrolled in this study, out of which 42 were enrolled in Part 1 and remaining 41 in Part 2.
Groups:
- Tanezumab 10 mcg/kg - Part 1: Single intravenous infusion of tanezumab 10 microgram/kilogram (mcg/kg) over 10 minutes on Day 1 during Part 1.
- Tanezumab 25 mcg/kg - Part 1: Single intravenous infusion of tanezumab 25 mcg/kg over 10 minutes on Day 1 during Part 1.
- Tanezumab 50 mcg/kg - Part 1: Single intravenous infusion of tanezumab 50 mcg/kg over 10 minutes on Day 1 during Part 1.
- Tanezumab 100 mcg/kg - Part 1: Single intravenous infusion of tanezumab 100 mcg/kg over 10 minutes on Day 1 during Part 1.
- Tanezumab 200 mcg/kg - Part 1: Single intravenous infusion of tanezumab 200 mcg/kg over 10 minutes on Day 1 during Part 1.
- Placebo - Part 1: Placebo matched to either of the single intravenous infusion over 10 minutes on Day 1 during Part 1.
- Tanezumab 10 mcg/kg - Part 2: Single intravenous infusion of tanezumab 10 mcg/kg over 10 minutes on Day 1 during Part 2.
- Tanezumab 25 mcg/kg - Part 2: Single intravenous infusion of tanezumab 25 mcg/kg over 10 minutes on Day 1 during Part 2.
- Tanezumab 50 mcg/kg - Part 2: Single intravenous infusion of tanezumab 50 mcg/kg over 10 minutes on Day 1 during Part 2.
- Tanezumab 100 mcg/kg - Part 2: Single intravenous infusion of tanezumab 100 mcg/kg over 10 minutes on Day 1 during Part 2.
- Placebo - Part 2: Placebo matched to either of the single intravenous infusion over 10 minutes on Day 1 during Part 2.
Period: Part 1
Arm/Group | Tanezumab 10 mcg/kg - Part 1 | Tanezumab 25 mcg/kg - Part 1 | Tanezumab 50 mcg/kg - Part 1 | Tanezumab 100 mcg/kg - Part 1 | Tanezumab 200 mcg/kg - Part 1 | Placebo - Part 1 | Tanezumab 10 mcg/kg - Part 2 | Tanezumab 25 mcg/kg - Part 2 | Tanezumab 50 mcg/kg - Part 2 | Tanezumab 100 mcg/kg - Part 2 | Placebo - Part 2
Started | 6 | 6 | 6 | 6 | 6 | 12 | 0 | 0 | 0 | 0 | 0
Completed | 6 | 6 | 6 | 6 | 6 | 12 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part 2
Arm/Group | Tanezumab 10 mcg/kg - Part 1 | Tanezumab 25 mcg/kg - Part 1 | Tanezumab 50 mcg/kg - Part 1 | Tanezumab 100 mcg/kg - Part 1 | Tanezumab 200 mcg/kg - Part 1 | Placebo - Part 1 | Tanezumab 10 mcg/kg - Part 2 | Tanezumab 25 mcg/kg - Part 2 | Tanezumab 50 mcg/kg - Part 2 | Tanezumab 100 mcg/kg - Part 2 | Placebo - Part 2
Started | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 9 | 9 | 10 | 4
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 9 | 9 | 9 | 9 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Tanezumab 10 mcg/kg: Single intravenous infusion of tanezumab 10 mcg/kg over 10 minutes on Day 1 during Part 1 and Part 2.
- Tanezumab 25 mcg/kg: Single intravenous infusion of tanezumab 25 mcg/kg over 10 minutes on Day 1 during Part 1 and Part 2.
- Tanezumab 50 mcg/kg: Single intravenous infusion of tanezumab 50 mcg/kg over 10 minutes on Day 1 during Part 1 and Part 2.
- Tanezumab 100 mcg/kg: Single intravenous infusion of tanezumab 100 mcg/kg over 10 minutes on Day 1 during Part 1 and Part 2.
- Tanezumab 200 mcg/kg: Single intravenous infusion of tanezumab 200 mcg/kg over 10 minutes on Day 1 during Part 1.
- Placebo: Placebo matched to either of the single intravenous infusion over 10 minutes on Day 1 during Part 1 and Part 2.
- Total: Total of all reporting groups
Arm/Group | Tanezumab 10 mcg/kg | Tanezumab 25 mcg/kg | Tanezumab 50 mcg/kg | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg | Placebo | Total
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 6 | 16 | 83
Age, Customized [Count of Participants; unit: Participants]
  36-45 Years | 0 | 0 | 0 | 1 | 0 | 0 | 1
  46-55 Years | 3 | 4 | 3 | 4 | 1 | 4 | 19
  56-65 Years | 12 | 11 | 10 | 9 | 5 | 11 | 58
  66-75 Years | 0 | 0 | 2 | 2 | 0 | 1 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 11 | 12 | 5 | 11 | 57
  Male | 5 | 7 | 4 | 4 | 1 | 5 | 26

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent: events between first dose of study drug and up to Day 1 through Day 120 (Part 1 and 2) were absent before treatment or that worsened relative to pretreatment state
Time Frame: Day 1 up to Day 92 for tanezumab 10, 25, 50 mcg/kg group and matching placebo group (Part 1, 2); Day 1 up to Day 120 for tanezumab 100 mcg/kg group and matching placebo group (Part 1, 2), 200 mcg/kg group and matching placebo group (Part 1)
Population: Safety analysis set included all participants who received single intravenous dose of study medication. It was planned to report combined data for Part 1 and 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Tanezumab 10 mcg/kg | Tanezumab 25 mcg/kg | Tanezumab 50 mcg/kg | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 6 | 16
Participants
  AEs | 9 | 4 | 9 | 8 | 6 | 13
  SAEs | 1 | 1 | 0 | 0 | 0 | 0

2. Primary Outcome: Hopkins Verbal Learning Test-Revised (HVLT-R) Total Score at Baseline
Description: The HVLT-R is an instrument used to measure verbal learning and memory (recognition and recall). It consists of 3 learning trials: free recall, delayed recall, and yes/no delayed recognition. The total recall score was the sum of 3 'free recall' learning trials, and reflects the participant's ability to learn. The total score ranges from 0 (no memory) to 36 (best memory). Higher score indicated best memory.
Time Frame: Baseline (Part 1 and Part 2)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mcg/kg | Tanezumab 25 mcg/kg | Tanezumab 50 mcg/kg | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 6 | 16
units on a scale | 27.1 (3.20) | 26.3 (4.48) | 24.1 (4.05) | 26.5 (4.29) | 27.2 (1.94) | 25.6 (5.14)

3. Primary Outcome: Hopkins Verbal Learning Test-Revised (HVLT-R) Total Score at Day 1
Description: as for outcome 2
Time Frame: Day 1 (Part 1 and 2)
Population: Safety analysis set included all participants who received single intravenous dose of study medication. Here, 'overall number of participants analyzed' signifies those who were evaluable for this measure. It was planned to report combined data for Part 1 and 2.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mcg/kg | Tanezumab 25 mcg/kg | Tanezumab 50 mcg/kg | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 12
units on a scale | 24.7 (2.42) | 23.2 (4.88) | 24.3 (2.07) | 27.3 (5.16) | 23.7 (2.58) | 23.5 (3.40)

4. Primary Outcome: Hopkins Verbal Learning Test-Revised (HVLT-R) Total Score at Day 4/5
Description: as for outcome 2
Time Frame: Day 4/5 (Part 1 and 2)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Tanezumab 10 mcg/kg: Single intravenous infusion of tanezumab 10 mcg/kg over 10 minutes on Day 1 during Part 1 and 2.
- Tanezumab 25 mcg/kg: Single intravenous infusion of tanezumab 25 mcg/kg over 10 minutes on Day 1 during Part 1 and 2.
- Tanezumab 50 mcg/kg: Single intravenous infusion of tanezumab 50 mcg/kg over 10 minutes on Day 1 during Part 1 and 2.
- Tanezumab 100 mcg/kg: Single intravenous infusion of tanezumab 100 mcg/kg over 10 minutes on Day 1 during Part 1 and 2.
- Placebo: Placebo matched to either of the single intravenous infusion over 10 minutes on Day 1 during Part 1 and 2.
Arm/Group | Tanezumab 10 mcg/kg | Tanezumab 25 mcg/kg | Tanezumab 50 mcg/kg | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 12
units on a scale | 27.7 (3.27) | 26.7 (3.01) | 27.0 (6.96) | 29.2 (3.92) | 26.0 (3.22) | 27.0 (3.36)

5. Primary Outcome: Hopkins Verbal Learning Test-Revised (HVLT-R) Total Score at Week 1
Description: as for outcome 2
Time Frame: Week 1 (Part 1 and Part 2)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mcg/kg | Tanezumab 25 mcg/kg | Tanezumab 50 mcg/kg | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 6 | 16
units on a scale | 26.7 (3.35) | 26.6 (4.81) | 25.4 (5.32) | 25.9 (5.15) | 26.8 (1.72) | 26.9 (4.15)

6. Primary Outcome: Hopkins Verbal Learning Test-Revised (HVLT-R) Total Score at Week 2
Description: as for outcome 2
Time Frame: Week 2 (Part 1 and Part 2)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mcg/kg | Tanezumab 25 mcg/kg | Tanezumab 50 mcg/kg | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 6 | 16
units on a scale | 27.0 (4.00) | 27.1 (4.32) | 25.7 (4.50) | 27.0 (5.98) | 25.5 (1.97) | 27.1 (3.60)

7. Primary Outcome: Hopkins Verbal Learning Test-Revised (HVLT-R) Total Score at Week 3
Description: as for outcome 2
Time Frame: Week 3 (Part 1 and 2)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Tanezumab 10 mcg/kg: Single intravenous infusion of tanezumab 10 mcg/kg over 10 minutes on Day 1 during Part 1.
- Tanezumab 25 mcg/kg: Single intravenous infusion of tanezumab 25 mcg/kg over 10 minutes on Day 1 during Part 1.
- Tanezumab 50 mcg/kg: Single intravenous infusion of tanezumab 50 mcg/kg over 10 minutes on Day 1 during Part 1.
- Tanezumab 100 mcg/kg: Single intravenous infusion of tanezumab 100 mcg/kg over 10 minutes on Day 1 during Part 1.
- Placebo: Placebo matched to either of the single intravenous infusion over 10 minutes on Day 1 during Part 1.
Arm/Group | Tanezumab 10 mcg/kg | Tanezumab 25 mcg/kg | Tanezumab 50 mcg/kg | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 12
units on a scale | 28.5 (5.75) | 30.3 (3.93) | 28.3 (4.27) | 31.2 (4.49) | 27.7 (2.07) | 27.8 (4.45)

8. Primary Outcome: Hopkins Verbal Learning Test-Revised (HVLT-R) Total Score at Week 4
Description: as for outcome 2
Time Frame: Week 4 (Part 1 and Part 2)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mcg/kg | Tanezumab 25 mcg/kg | Tanezumab 50 mcg/kg | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 6 | 16
units on a scale | 28.5 (3.60) | 26.4 (5.45) | 27.2 (4.02) | 27.6 (4.86) | 27.0 (3.58) | 26.9 (4.75)

9. Primary Outcome: Hopkins Verbal Learning Test-Revised (HVLT-R) Total Score at Week 13
Description: as for outcome 2
Time Frame: Week 13 (Part 1 and Part 2)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mcg/kg | Tanezumab 25 mcg/kg | Tanezumab 50 mcg/kg | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 6 | 16
units on a scale | 28.5 (4.16) | 26.8 (5.23) | 27.3 (3.92) | 28.8 (5.87) | 23.8 (1.83) | 26.0 (4.32)

10. Primary Outcome: Hopkins Verbal Learning Test-Revised (HVLT-R) Total Score at Week 17
Description: as for outcome 2
Time Frame: Week 17 (Part 1 and Part 2)
Population: Safety analysis set included all participants who received single intravenous dose of study medication. Week 17 analyses was performed only for treatment arms Tanezumab 100 mcg/kg, 200 mcg/kg and Placebo as per analysis plan. It was planned to report combined data for Part 1 and 2.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg | Placebo
Number analyzed (Participants) | 16 | 6 | 16
units on a scale | 29.3 (5.27) | 27.3 (2.07) | 28.9 (3.72)

11. Primary Outcome: Change From Baseline in Visual Analogue Scale (VAS) Score For Current Index Knee Pain at Week 1
Description: VAS assesses participant responses from 0 to 100 (0 = none to 100 = extreme) with 101 point resolution for measuring pain intensity. Higher score indicated greater pain intensity. VAS for current index knee pain was recorded on the electronic diary.
Time Frame: Baseline, Week 1 (Part 1 and 2)
Population: Full Analysis Set (FAS) included all participants who had received full single intravenous dose of study medication and had at least one entry of electronic diary in both pre and post treatments. Here, 'overall number of participants analyzed' signifies those who were evaluable for this measure. It was planned to report combined data for Part 1 and 2.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mcg/kg | Tanezumab 25 mcg/kg | Tanezumab 50 mcg/kg | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 6 | 14
units on a scale
  Baseline | 66.5 (22.61) | 64.5 (12.49) | 67.9 (8.41) | 65.0 (13.77) | 69.7 (9.27) | 62.3 (18.86)
  Change at Week 1 | -13.9 (17.75) | -29.7 (22.10) | -15.0 (19.96) | -25.2 (20.35) | -46.6 (21.62) | -10.1 (9.31)
Statistical Analysis 1: Comparison: Tanezumab 10 mcg/kg vs Placebo; Mixed Model for Repeated Measures analyses included fixed effects of treatment, week, treatment by week, part, and baseline values; Test type: Superiority or Other; Least Square Mean Difference = -2.0, 95% CI 2-sided [-17.8 to 13.8], Standard Error of Mean 7.98
Statistical Analysis 2: Comparison: Tanezumab 25 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -18.5, 95% CI 2-sided [-34.3 to -2.8], Standard Error of Mean 7.98
Statistical Analysis 3: Comparison: Tanezumab 50 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -2.7, 95% CI 2-sided [-18.5 to 13.1], Standard Error of Mean 7.99
Statistical Analysis 4: Comparison: Tanezumab 100 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -13.8, 95% CI 2-sided [-29.4 to 1.8], Standard Error of Mean 7.88
Statistical Analysis 5: Comparison: Tanezumab 200 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -34.5, 95% CI 2-sided [-55.2 to -13.7], Standard Error of Mean 10.48

12. Primary Outcome: Change From Baseline in Visual Analogue Scale (VAS) Score For Current Index Knee Pain at Week 2
Description: as for outcome 11
Time Frame: Baseline, Week 2 (Part 1 and 2)
Population: FAS included all participants who had received full single intravenous dose of study medication and had at least one entry of electronic diary in both pre and post treatments. Here, 'overall number of participants analyzed' signifies those who were evaluable for this measure. It was planned to report combined data for Part 1 and 2.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mcg/kg | Tanezumab 25 mcg/kg | Tanezumab 50 mcg/kg | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 6 | 14
units on a scale | -18.6 (19.82) | -29.3 (25.09) | -11.3 (19.89) | -25.5 (20.48) | -25.1 (26.23) | -13.2 (16.20)
Statistical Analysis 1: Comparison: Tanezumab 10 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -3.6, 95% CI 2-sided [-19.4 to 12.2], Standard Error of Mean 7.98
Statistical Analysis 2: Comparison: Tanezumab 25 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -15.0, 95% CI 2-sided [-30.8 to 0.8], Standard Error of Mean 7.98
Statistical Analysis 3: Comparison: Tanezumab 50 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = 4.1, 95% CI 2-sided [-11.7 to 19.9], Standard Error of Mean 7.99
Statistical Analysis 4: Comparison: Tanezumab 100 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -11.0, 95% CI 2-sided [-26.6 to 4.6], Standard Error of Mean 7.88
Statistical Analysis 5: Comparison: Tanezumab 200 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -9.8, 95% CI 2-sided [-30.5 to 10.9], Standard Error of Mean 10.48

13. Primary Outcome: Change From Baseline in Visual Analogue Scale (VAS) Score For Current Index Knee Pain at Week 3
Description: as for outcome 11
Time Frame: Baseline, Week 3 (Part 1 and 2)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mcg/kg | Tanezumab 25 mcg/kg | Tanezumab 50 mcg/kg | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 6 | 14
units on a scale | -21.7 (21.33) | -35.9 (24.58) | -15.3 (22.49) | -27.0 (18.19) | -23.0 (27.44) | -16.3 (20.41)
Statistical Analysis 1: Comparison: Tanezumab 10 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -3.6, 95% CI 2-sided [-19.4 to 12.2], Standard Error of Mean 7.98
Statistical Analysis 2: Comparison: Tanezumab 25 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -18.5, 95% CI 2-sided [-34.3 to -2.8], Standard Error of Mean 7.98
Statistical Analysis 3: Comparison: Tanezumab 50 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = 3.2, 95% CI 2-sided [-12.6 to 19.0], Standard Error of Mean 7.99
Statistical Analysis 4: Comparison: Tanezumab 100 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -9.4, 95% CI 2-sided [-25.0 to 6.2], Standard Error of Mean 7.88
Statistical Analysis 5: Comparison: Tanezumab 200 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -4.6, 95% CI 2-sided [-25.4 to 16.1], Standard Error of Mean 10.48

14. Primary Outcome: Change From Baseline in Visual Analogue Scale (VAS) Score For Current Index Knee Pain at Week 4
Description: as for outcome 11
Time Frame: Baseline, Week 4 (Part 1 and 2)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mcg/kg | Tanezumab 25 mcg/kg | Tanezumab 50 mcg/kg | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 6 | 14
units on a scale | -22.3 (21.30) | -37.1 (24.96) | -21.8 (21.41) | -30.6 (18.15) | -46.0 (17.47) | -18.2 (21.73)
Statistical Analysis 1: Comparison: Tanezumab 10 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -2.3, 95% CI 2-sided [-18.1 to 13.5], Standard Error of Mean 7.98
Statistical Analysis 2: Comparison: Tanezumab 25 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -17.8, 95% CI 2-sided [-33.6 to -2.1], Standard Error of Mean 7.98
Statistical Analysis 3: Comparison: Tanezumab 50 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -1.4, 95% CI 2-sided [-17.2 to 14.4], Standard Error of Mean 7.99
Statistical Analysis 4: Comparison: Tanezumab 100 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -11.2, 95% CI 2-sided [-26.7 to 4.4], Standard Error of Mean 7.88
Statistical Analysis 5: Comparison: Tanezumab 200 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -25.8, 95% CI 2-sided [-46.5 to -5.0], Standard Error of Mean 10.48

15. Primary Outcome: Change From Baseline in Visual Analogue Scale (VAS) Score For Current Index Knee Pain at Week 5
Description: as for outcome 11
Time Frame: Baseline, Week 5 (Part 1 and 2)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mcg/kg | Tanezumab 25 mcg/kg | Tanezumab 50 mcg/kg | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 6 | 14
units on a scale | -22.3 (22.25) | -38.0 (23.44) | -27.2 (24.90) | -33.8 (19.02) | -50.7 (15.36) | -19.8 (23.07)
Statistical Analysis 1: Comparison: Tanezumab 10 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -0.8, 95% CI 2-sided [-16.6 to 15.0], Standard Error of Mean 7.98
Statistical Analysis 2: Comparison: Tanezumab 25 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -17.1, 95% CI 2-sided [-32.8 to -1.3], Standard Error of Mean 7.98
Statistical Analysis 3: Comparison: Tanezumab 50 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -5.2, 95% CI 2-sided [-21.0 to 10.6], Standard Error of Mean 7.99
Statistical Analysis 4: Comparison: Tanezumab 100 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -12.7, 95% CI 2-sided [-28.3 to 2.9], Standard Error of Mean 7.88
Statistical Analysis 5: Comparison: Tanezumab 200 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -28.9, 95% CI 2-sided [-49.6 to -8.2], Standard Error of Mean 10.48

16. Primary Outcome: Change From Baseline In Visual Analogue Scale (VAS) Score For Current Index Knee Pain at Week 6
Description: as for outcome 11
Time Frame: Baseline, Week 6 (Part 1 and 2)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mcg/kg | Tanezumab 25 mcg/kg | Tanezumab 50 mcg/kg | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 6 | 14
units on a scale | -22.2 (23.49) | -39.8 (24.56) | -27.7 (24.73) | -33.2 (19.14) | -51.4 (17.13) | -19.5 (24.01)
Statistical Analysis 1: Comparison: Tanezumab 10 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -1.0, 95% CI 2-sided [-16.8 to 14.8], Standard Error of Mean 7.98
Statistical Analysis 2: Comparison: Tanezumab 25 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -19.3, 95% CI 2-sided [-35.0 to -3.5], Standard Error of Mean 7.98
Statistical Analysis 3: Comparison: Tanezumab 50 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -6.0, 95% CI 2-sided [-21.8 to 9.8], Standard Error of Mean 7.99
Statistical Analysis 4: Comparison: Tanezumab 100 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -12.4, 95% CI 2-sided [-28.0 to 3.2], Standard Error of Mean 7.88
Statistical Analysis 5: Comparison: Tanezumab 200 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -29.9, 95% CI 2-sided [-50.6 to -9.1], Standard Error of Mean 10.48

17. Primary Outcome: Change From Baseline In Visual Analogue Scale (VAS) Score For Current Index Knee Pain at Week 7
Description: VAS assesses participant responses from 0 to 100 (0 = none to 10 0= extreme) with 101 point resolution for measuring pain intensity. Higher score indicated greater pain intensity. VAS for current index knee pain was recorded on the electronic diary.
Time Frame: Baseline, Week 7 (Part 1 and 2)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mcg/kg | Tanezumab 25 mcg/kg | Tanezumab 50 mcg/kg | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 6 | 14
units on a scale | -18.7 (23.34) | -41.2 (24.30) | -28.5 (24.77) | -34.3 (18.43) | -47.9 (14.28) | -20.8 (23.62)
Statistical Analysis 1: Comparison: Tanezumab 10 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = 3.9, 95% CI 2-sided [-11.9 to 19.7], Standard Error of Mean 7.98
Statistical Analysis 2: Comparison: Tanezumab 25 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -19.3, 95% CI 2-sided [-35.1 to -3.6], Standard Error of Mean 7.98
Statistical Analysis 3: Comparison: Tanezumab 50 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -5.5, 95% CI 2-sided [-21.3 to 10.3], Standard Error of Mean 7.99
Statistical Analysis 4: Comparison: Tanezumab 100 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -12.2, 95% CI 2-sided [-27.8 to 3.4], Standard Error of Mean 7.88
Statistical Analysis 5: Comparison: Tanezumab 200 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -25.0, 95% CI 2-sided [-45.8 to -4.3], Standard Error of Mean 10.48

18. Primary Outcome: Change From Baseline In Visual Analogue Scale (VAS) Score For Current Index Knee Pain at Week 8
Description: as for outcome 11
Time Frame: Baseline, Week 8 (Part 1 and 2)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mcg/kg | Tanezumab 25 mcg/kg | Tanezumab 50 mcg/kg | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 6 | 14
units on a scale | -17.8 (23.35) | -39.8 (24.94) | -27.6 (24.86) | -34.3 (17.98) | -48.2 (16.18) | -22.7 (23.67)
Statistical Analysis 1: Comparison: Tanezumab 10 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = 6.7, 95% CI 2-sided [-9.1 to 22.5], Standard Error of Mean 7.98
Statistical Analysis 2: Comparison: Tanezumab 25 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -16.0, 95% CI 2-sided [-31.7 to -0.2], Standard Error of Mean 7.98
Statistical Analysis 3: Comparison: Tanezumab 50 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -2.6, 95% CI 2-sided [-18.5 to 13.2], Standard Error of Mean 7.99
Statistical Analysis 4: Comparison: Tanezumab 100 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -10.3, 95% CI 2-sided [-25.9 to 5.3], Standard Error of Mean 7.88
Statistical Analysis 5: Comparison: Tanezumab 200 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -23.5, 95% CI 2-sided [-44.2 to -2.7], Standard Error of Mean 10.48

19. Primary Outcome: Change From Baseline in Visual Analogue Scale (VAS) Score For Current Index Knee Pain at Week 9
Description: as for outcome 11
Time Frame: Baseline, Week 9 (Part 1 and 2)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mcg/kg | Tanezumab 25 mcg/kg | Tanezumab 50 mcg/kg | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 6 | 14
units on a scale | -16.4 (23.80) | -41.2 (26.62) | -26.5 (23.77) | -33.4 (19.60) | -47.6 (11.81) | -25.8 (24.77)
Statistical Analysis 1: Comparison: Tanezumab 10 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = 11.2, 95% CI 2-sided [-4.6 to 27.0], Standard Error of Mean 7.98
Statistical Analysis 2: Comparison: Tanezumab 25 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -14.2, 95% CI 2-sided [-30.0 to 1.5], Standard Error of Mean 7.98
Statistical Analysis 3: Comparison: Tanezumab 50 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = 1.5, 95% CI 2-sided [-14.3 to 17.3], Standard Error of Mean 7.99
Statistical Analysis 4: Comparison: Tanezumab 100 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -6.3, 95% CI 2-sided [-21.9 to 9.3], Standard Error of Mean 7.88
Statistical Analysis 5: Comparison: Tanezumab 200 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -19.8, 95% CI 2-sided [-40.5 to 1.0], Standard Error of Mean 10.48

20. Primary Outcome: Change From Baseline in Visual Analogue Scale (VAS) Score For Current Index Knee Pain at Week 10
Description: as for outcome 11
Time Frame: Baseline, Week 10 (Part 1 and 2)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mcg/kg | Tanezumab 25 mcg/kg | Tanezumab 50 mcg/kg | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 6 | 14
units on a scale | -15.5 (20.94) | -39.9 (28.09) | -25.6 (23.44) | -31.2 (18.94) | -41.2 (14.35) | -24.6 (23.50)
Statistical Analysis 1: Comparison: Tanezumab 10 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = 10.8, 95% CI 2-sided [-5.0 to 26.6], Standard Error of Mean 7.98
Statistical Analysis 2: Comparison: Tanezumab 25 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -14.2, 95% CI 2-sided [-30.0 to 1.6], Standard Error of Mean 7.98
Statistical Analysis 3: Comparison: Tanezumab 50 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = 1.2, 95% CI 2-sided [-14.6 to 17.0], Standard Error of Mean 7.99
Statistical Analysis 4: Comparison: Tanezumab 100 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -5.4, 95% CI 2-sided [-21.0 to 10.2], Standard Error of Mean 7.88
Statistical Analysis 5: Comparison: Tanezumab 200 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -14.6, 95% CI 2-sided [-35.3 to 6.2], Standard Error of Mean 10.48

21. Primary Outcome: Change From Baseline in Visual Analogue Scale (VAS) Score For Current Index Knee Pain at Week 11
Description: as for outcome 11
Time Frame: Baseline, Week 11 (Part 1 and 2)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mcg/kg | Tanezumab 25 mcg/kg | Tanezumab 50 mcg/kg | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 6 | 14
units on a scale | -17.1 (19.92) | -38.0 (25.04) | -25.4 (23.41) | -30.6 (17.75) | -41.4 (20.24) | -25.7 (23.27)
Statistical Analysis 1: Comparison: Tanezumab 10 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = 10.3, 95% CI 2-sided [-5.5 to 26.1], Standard Error of Mean 7.98
Statistical Analysis 2: Comparison: Tanezumab 25 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -11.3, 95% CI 2-sided [-27.0 to 4.5], Standard Error of Mean 7.98
Statistical Analysis 3: Comparison: Tanezumab 50 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = 2.5, 95% CI 2-sided [-13.3 to 18.3], Standard Error of Mean 7.99
Statistical Analysis 4: Comparison: Tanezumab 100 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -3.7, 95% CI 2-sided [-19.2 to 11.9], Standard Error of Mean 7.88
Statistical Analysis 5: Comparison: Tanezumab 200 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -13.7, 95% CI 2-sided [-34.4 to 7.0], Standard Error of Mean 10.48

22. Primary Outcome: Change From Baseline in Visual Analogue Scale (VAS) Score For Current Index Knee Pain at Week 12
Description: as for outcome 11
Time Frame: Baseline, Week 12 (Part 1 and 2)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mcg/kg | Tanezumab 25 mcg/kg | Tanezumab 50 mcg/kg | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 6 | 14
units on a scale | -16.2 (21.34) | -34.7 (24.93) | -25.8 (23.06) | -30.3 (18.56) | -40.3 (22.88) | -25.4 (25.76)
Statistical Analysis 1: Comparison: Tanezumab 10 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Mean Square Difference = 11.0, 95% CI 2-sided [-4.8 to 26.8], Standard Error of Mean 7.98
Statistical Analysis 2: Comparison: Tanezumab 25 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Mean Square Difference = -8.1, 95% CI 2-sided [-23.9 to 7.6], Standard Error of Mean 7.98
Statistical Analysis 3: Comparison: Tanezumab 50 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Mean Square Difference = 1.8, 95% CI 2-sided [-14.0 to 17.6], Standard Error of Mean 7.99
Statistical Analysis 4: Comparison: Tanezumab 100 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Mean Square Difference = -3.6, 95% CI 2-sided [-19.2 to 12.0], Standard Error of Mean 7.88
Statistical Analysis 5: Comparison: Tanezumab 200 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Mean Square Difference = -12.8, 95% CI 2-sided [-33.5 to 8.0], Standard Error of Mean 10.48

23. Primary Outcome: Change From Baseline in Visual Analogue Scale (VAS) Score For Current Index Knee Pain at Week 13
Description: as for outcome 11
Time Frame: Baseline, Week 13 (Part 1 and 2)
Population: FAS included all participants who had received full single intravenous dose of study medication and had at least one entry of electronic diary in both pre and post treatments. Here, 'overall number of participants analyzed' signify those who were evaluable for this measure. It was planned to report combined data for Part 1 and 2.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mcg/kg | Tanezumab 25 mcg/kg | Tanezumab 50 mcg/kg | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 6 | 14
units on a scale | -15.8 (21.64) | -32.0 (25.89) | -23.0 (22.15) | -32.0 (19.67) | -31.6 (28.83) | -25.4 (26.56)
Statistical Analysis 1: Comparison: Tanezumab 10 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Mean Square Difference = 11.4, 95% CI 2-sided [-4.4 to 27.2], Standard Error of Mean 7.98
Statistical Analysis 2: Comparison: Tanezumab 25 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Mean Square Difference = -5.4, 95% CI 2-sided [-21.2 to 10.3], Standard Error of Mean 7.98
Statistical Analysis 3: Comparison: Tanezumab 50 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Mean Square Difference = 4.6, 95% CI 2-sided [-11.2 to 20.4], Standard Error of Mean 7.99
Statistical Analysis 4: Comparison: Tanezumab 100 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Mean Square Difference = -4.7, 95% CI 2-sided [-20.3 to 10.9], Standard Error of Mean 7.89
Statistical Analysis 5: Comparison: Tanezumab 200 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Mean Square Difference = -4.1, 95% CI 2-sided [-24.9 to 16.6], Standard Error of Mean 10.48

24. Primary Outcome: Change From Baseline Visual Analogue Scale (VAS) Score For Index Knee Pain in the Past 24 Hours at Week 1
Description: VAS assesses participant responses from 0 to 100 (0 = none to 100 = extreme) with 101 point resolution for measuring pain intensity. Higher score indicated greater pain intensity. VAS for index knee pain in the past 24 hours was recorded on the electronic diary.
Time Frame: Baseline, Week 1 (Part 1 and 2)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mcg/kg | Tanezumab 25 mcg/kg | Tanezumab 50 mcg/kg | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 6 | 14
units on a scale
  Baseline | 75.4 (9.32) | 67.3 (11.24) | 70.6 (8.63) | 67.8 (10.70) | 69.0 (11.37) | 68.0 (14.27)
  Change at Week 1 | -17.3 (19.59) | -29.8 (22.13) | -15.7 (19.33) | -26.4 (20.78) | -45.2 (17.49) | -10.2 (10.83)
Statistical Analysis 1: Comparison: Tanezumab 10 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Mean Square Difference = -4.2, 95% CI 2-sided [-20.7 to 12.3], Standard Error of Mean 8.33
Statistical Analysis 2: Comparison: Tanezumab 25 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Mean Square Difference = -19.3, 95% CI 2-sided [-35.6 to -3.0], Standard Error of Mean 8.25
Statistical Analysis 3: Comparison: Tanezumab 50 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Mean Square Difference = -4.2, 95% CI 2-sided [-20.5 to 12.1], Standard Error of Mean 8.25
Statistical Analysis 4: Comparison: Tanezumab 100 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Mean Square Difference = -15.8, 95% CI 2-sided [-31.9 to 0.3], Standard Error of Mean 8.14
Statistical Analysis 5: Comparison: Tanezumab 200 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Mean Square Difference = -35.1, 95% CI 2-sided [-56.4 to -13.8], Standard Error of Mean 10.75

25. Primary Outcome: Change From Baseline in Visual Analogue Scale (VAS) Score For Index Knee Pain in the Past 24 Hours at Week 2
Description: as for outcome 24
Time Frame: Baseline, Week 2 (Part 1 and 2)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mcg/kg | Tanezumab 25 mcg/kg | Tanezumab 50 mcg/kg | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 6 | 14
units on a scale | -20.6 (18.94) | -29.9 (26.26) | -11.5 (19.62) | -26.5 (19.31) | -24.4 (27.09) | -13.0 (17.53)
Statistical Analysis 1: Comparison: Tanezumab 10 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -4.7, 95% CI 2-sided [-21.2 to 11.8], Standard Error of Mean 8.33
Statistical Analysis 2: Comparison: Tanezumab 25 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -16.7, 95% CI 2-sided [-33.0 to -0.4], Standard Error of Mean 8.25
Statistical Analysis 3: Comparison: Tanezumab 50 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = 2.8, 95% CI 2-sided [-13.5 to 19.1], Standard Error of Mean 8.25
Statistical Analysis 4: Comparison: Tanezumab 100 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -13.1, 95% CI 2-sided [-29.2 to 3.0], Standard Error of Mean 8.14
Statistical Analysis 5: Comparison: Tanezumab 200 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -11.5, 95% CI 2-sided [-32.8 to 9.7], Standard Error of Mean 10.75

26. Primary Outcome: Change From Baseline in Visual Analogue Scale (VAS) Score For Index Knee Pain in the Past 24 Hours at Week 3
Description: as for outcome 24
Time Frame: Baseline, Week 3 (Part 1 and 2)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mcg/kg | Tanezumab 25 mcg/kg | Tanezumab 50 mcg/kg | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 6 | 14
units on a scale | -25.9 (19.75) | -36.2 (25.06) | -16.5 (22.85) | -28.0 (18.82) | -21.2 (28.87) | -16.6 (21.73)
Statistical Analysis 1: Comparison: Tanezumab 10 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -6.4, 95% CI 2-sided [-22.9 to 10.1], Standard Error of Mean 8.33
Statistical Analysis 2: Comparison: Tanezumab 25 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -19.4, 95% CI 2-sided [-35.7 to -3.1], Standard Error of Mean 8.25
Statistical Analysis 3: Comparison: Tanezumab 50 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = 1.3, 95% CI 2-sided [-15.0 to 17.6], Standard Error of Mean 8.25
Statistical Analysis 4: Comparison: Tanezumab 100 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -11.0, 95% CI 2-sided [-27.1 to 5.1], Standard Error of Mean 8.14
Statistical Analysis 5: Comparison: Tanezumab 200 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -4.8, 95% CI 2-sided [-26.0 to 16.5], Standard Error of Mean 10.75

27. Primary Outcome: Change From Baseline in Visual Analogue Scale (VAS) Score For Index Knee Pain in the Past 24 Hours at Week 4
Description: as for outcome 24
Time Frame: Baseline, Week 4 (Part 1 and 2)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mcg/kg | Tanezumab 25 mcg/kg | Tanezumab 50 mcg/kg | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 6 | 14
units on a scale | -25.5 (20.07) | -37.9 (26.37) | -23.4 (22.07) | -32.3 (18.00) | -45.4 (18.10) | -18.0 (23.39)
Statistical Analysis 1: Comparison: Tanezumab 10 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -4.6, 95% CI 2-sided [-21.1 to 11.9], Standard Error of Mean 8.33
Statistical Analysis 2: Comparison: Tanezumab 25 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -19.6, 95% CI 2-sided [-35.9 to -3.3], Standard Error of Mean 8.25
Statistical Analysis 3: Comparison: Tanezumab 50 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -4.1, 95% CI 2-sided [-20.4 to 12.2], Standard Error of Mean 8.25
Statistical Analysis 4: Comparison: Tanezumab 100 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -13.8, 95% CI 2-sided [-30.0 to 2.3], Standard Error of Mean 8.14
Statistical Analysis 5: Comparison: Tanezumab 200 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -27.5, 95% CI 2-sided [-48.8 to -6.2], Standard Error of Mean 10.75

28. Primary Outcome: Change From Baseline in Visual Analogue Scale (VAS) Score For Index Knee Pain in The Past 24 Hours at Week 5
Description: as for outcome 24
Time Frame: Baseline, Week 5 (Part 1 and 2)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mcg/kg | Tanezumab 25 mcg/kg | Tanezumab 50 mcg/kg | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 6 | 14
units on a scale | -24.3 (22.64) | -38.1 (25.13) | -28.7 (24.64) | -35.4 (19.03) | -50.8 (15.62) | -18.3 (25.31)
Statistical Analysis 1: Comparison: Tanezumab 10 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -3.1, 95% CI 2-sided [-19.6 to 13.4], Standard Error of Mean 8.33
Statistical Analysis 2: Comparison: Tanezumab 25 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -19.5, 95% CI 2-sided [-35.8 to -3.1], Standard Error of Mean 8.25
Statistical Analysis 3: Comparison: Tanezumab 50 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -9.1, 95% CI 2-sided [-25.4 to 7.2], Standard Error of Mean 8.25
Statistical Analysis 4: Comparison: Tanezumab 100 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -16.6, 95% CI 2-sided [-32.8 to -0.5], Standard Error of Mean 8.14
Statistical Analysis 5: Comparison: Tanezumab 200 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -32.6, 95% CI 2-sided [-53.9 to -11.4], Standard Error of Mean 10.75

29. Primary Outcome: Change From Baseline in Visual Analogue Scale (VAS) Score For Index Knee Pain in the Past 24 Hours at Week 6
Description: as for outcome 24
Time Frame: Baseline, Week 6 (Part 1 and 2)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mcg/kg | Tanezumab 25 mcg/kg | Tanezumab 50 mcg/kg | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 6 | 14
units on a scale | -24.7 (24.85) | -40.0 (25.22) | -28.9 (25.30) | -34.1 (17.86) | -50.6 (16.59) | -18.2 (26.35)
Statistical Analysis 1: Comparison: Tanezumab 10 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -3.6, 95% CI 2-sided [-20.1 to 12.9], Standard Error of Mean 8.33
Statistical Analysis 2: Comparison: Tanezumab 25 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -21.5, 95% CI 2-sided [-37.9 to -5.2], Standard Error of Mean 8.25
Statistical Analysis 3: Comparison: Tanezumab 50 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -9.4, 95% CI 2-sided [-25.7 to 6.9], Standard Error of Mean 8.25
Statistical Analysis 4: Comparison: Tanezumab 100 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -15.4, 95% CI 2-sided [-31.5 to 0.7], Standard Error of Mean 8.14
Statistical Analysis 5: Comparison: Tanezumab 200 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -32.5, 95% CI 2-sided [-53.7 to -11.2], Standard Error of Mean 10.75

30. Primary Outcome: Change From Baseline in Visual Analogue Scale (VAS) Score For Index Knee Pain in the Past 24 Hours at Week 7
Description: as for outcome 24
Time Frame: Baseline, Week 7 (Part 1 and 2)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mcg/kg | Tanezumab 25 mcg/kg | Tanezumab 50 mcg/kg | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 6 | 14
units on a scale | -22.9 (23.08) | -41.1 (24.78) | -28.7 (25.90) | -36.1 (18.19) | -46.3 (14.37) | -19.6 (26.21)
Statistical Analysis 1: Comparison: Tanezumab 10 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -0.5, 95% CI 2-sided [-17.0 to 16.0], Standard Error of Mean 8.33
Statistical Analysis 2: Comparison: Tanezumab 25 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -21.3, 95% CI 2-sided [-37.6 to -4.9], Standard Error of Mean 8.25
Statistical Analysis 3: Comparison: Tanezumab 50 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -7.8, 95% CI 2-sided [-24.1 to 8.5], Standard Error of Mean 8.25
Statistical Analysis 4: Comparison: Tanezumab 100 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -16.1, 95% CI 2-sided [-32.2 to 0.0], Standard Error of Mean 8.14
Statistical Analysis 5: Comparison: Tanezumab 200 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -26.8, 95% CI 2-sided [-48.1 to -5.5], Standard Error of Mean 10.75

31. Primary Outcome: Change From Baseline in Visual Analogue Scale (VAS) Score For Index Knee Pain in the Past 24 Hours at Week 8
Description: as for outcome 24
Time Frame: Baseline, Week 8 (Part 1 and 2)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mcg/kg | Tanezumab 25 mcg/kg | Tanezumab 50 mcg/kg | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 6 | 14
units on a scale | -21.2 (23.17) | -40.8 (25.93) | -28.7 (25.65) | -36.4 (18.34) | -46.7 (16.38) | -22.0 (25.87)
Statistical Analysis 1: Comparison: Tanezumab 10 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = 3.7, 95% CI 2-sided [-12.8 to 20.2], Standard Error of Mean 8.33
Statistical Analysis 2: Comparison: Tanezumab 25 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -18.5, 95% CI 2-sided [-34.8 to -2.2], Standard Error of Mean 8.25
Statistical Analysis 3: Comparison: Tanezumab 50 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -5.3, 95% CI 2-sided [-21.7 to 11.0], Standard Error of Mean 8.25
Statistical Analysis 4: Comparison: Tanezumab 100 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -14.0, 95% CI 2-sided [-30.1 to 2.1], Standard Error of Mean 8.14
Statistical Analysis 5: Comparison: Tanezumab 200 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -24.8, 95% CI 2-sided [-46.0 to -3.5], Standard Error of Mean 10.75

32. Primary Outcome: Change From Baseline in Visual Analogue Scale (VAS) Score For Index Knee Pain in the Past 24 Hours at Week 9
Description: as for outcome 24
Time Frame: Baseline, Week 9 (Part 1 and 2)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mcg/kg | Tanezumab 25 mcg/kg | Tanezumab 50 mcg/kg | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 6 | 14
units on a scale | -19.2 (22.76) | -41.3 (27.52) | -27.1 (24.72) | -35.2 (19.54) | -46.0 (11.44) | -25.4 (25.41)
Statistical Analysis 1: Comparison: Tanezumab 10 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = 9.0, 95% CI 2-sided [-7.5 to 25.5], Standard Error of Mean 8.33
Statistical Analysis 2: Comparison: Tanezumab 25 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -15.7, 95% CI 2-sided [-32.0 to 0.6], Standard Error of Mean 8.25
Statistical Analysis 3: Comparison: Tanezumab 50 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -0.4, 95% CI 2-sided [-16.7 to 15.9], Standard Error of Mean 8.25
Statistical Analysis 4: Comparison: Tanezumab 100 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -9.4, 95% CI 2-sided [-25.5 to 6.7], Standard Error of Mean 8.14
Statistical Analysis 5: Comparison: Tanezumab 200 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -20.8, 95% CI 2-sided [-42.0 to 0.5], Standard Error of Mean 10.75

33. Primary Outcome: Change From Baseline in Visual Analogue Scale (VAS) Score For Index Knee Pain in the Past 24 Hours at Week 10
Description: as for outcome 24
Time Frame: Baseline, Week 10 (Part 1 and 2)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mcg/kg | Tanezumab 25 mcg/kg | Tanezumab 50 mcg/kg | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 6 | 14
units on a scale | -18.7 (20.60) | -40.6 (28.43) | -26.1 (24.58) | -32.7 (18.45) | -40.6 (13.00) | -24.0 (25.24)
Statistical Analysis 1: Comparison: Tanezumab 10 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = 8.1, 95% CI 2-sided [-8.4 to 24.6], Standard Error of Mean 8.33
Statistical Analysis 2: Comparison: Tanezumab 25 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -16.3, 95% CI 2-sided [-32.6 to 0.0], Standard Error of Mean 8.25
Statistical Analysis 3: Comparison: Tanezumab 50 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -0.8, 95% CI 2-sided [-17.1 to 15.5], Standard Error of Mean 8.25
Statistical Analysis 4: Comparison: Tanezumab 100 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -8.3, 95% CI 2-sided [-24.4 to 7.8], Standard Error of Mean 8.14
Statistical Analysis 5: Comparison: Tanezumab 200 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -16.7, 95% CI 2-sided [-38.0 to 4.5], Standard Error of Mean 10.75

34. Primary Outcome: Change From Baseline in Visual Analogue Scale (VAS) Score For Index Knee Pain in the Past 24 Hours at Week 11
Description: as for outcome 24
Time Frame: Baseline, Week 11 (Part 1 and 2)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mcg/kg | Tanezumab 25 mcg/kg | Tanezumab 50 mcg/kg | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 6 | 14
units on a scale | -18.9 (18.93) | -38.0 (25.76) | -25.7 (24.08) | -32.8 (17.99) | -40.5 (19.64) | -24.8 (24.72)
Statistical Analysis 1: Comparison: Tanezumab 10 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = 8.8, 95% CI 2-sided [-7.7 to 25.3], Standard Error of Mean 8.33
Statistical Analysis 2: Comparison: Tanezumab 25 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -12.9, 95% CI 2-sided [-29.2 to 3.5], Standard Error of Mean 8.25
Statistical Analysis 3: Comparison: Tanezumab 50 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = 0.5, 95% CI 2-sided [-15.8 to 16.8], Standard Error of Mean 8.25
Statistical Analysis 4: Comparison: Tanezumab 100 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -7.5, 95% CI 2-sided [-23.6 to 8.6], Standard Error of Mean 8.14
Statistical Analysis 5: Comparison: Tanezumab 200 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -15.7, 95% CI 2-sided [-37.0 to 5.5], Standard Error of Mean 10.75

35. Primary Outcome: Change From Baseline in Visual Analogue Scale (VAS) Score For Index Knee Pain in the Past 24 Hours at Week 12
Description: as for outcome 24
Time Frame: Baseline, Week 12 (Part 1 and 2)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mcg/kg | Tanezumab 25 mcg/kg | Tanezumab 50 mcg/kg | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 6 | 14
units on a scale | -17.9 (19.78) | -35.1 (24.85) | -25.9 (24.09) | -32.3 (19.04) | -39.8 (21.06) | -24.1 (26.15)
Statistical Analysis 1: Comparison: Tanezumab 10 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = 9.0, 95% CI 2-sided [-7.4 to 25.5], Standard Error of Mean 8.33
Statistical Analysis 2: Comparison: Tanezumab 25 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -10.8, 95% CI 2-sided [-27.1 to 5.5], Standard Error of Mean 8.25
Statistical Analysis 3: Comparison: Tanezumab 50 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -0.6, 95% CI 2-sided [-16.9 to 15.7], Standard Error of Mean 8.25
Statistical Analysis 4: Comparison: Tanezumab 100 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -7.8, 95% CI 2-sided [-23.9 to 8.4], Standard Error of Mean 8.14
Statistical Analysis 5: Comparison: Tanezumab 200 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -15.8, 95% CI 2-sided [-37.1 to 5.4], Standard Error of Mean 10.75

36. Primary Outcome: Change From Baseline in Visual Analogue Scale (VAS) Score For Index Knee Pain in the Past 24 Hours at Week 13
Description: as for outcome 24
Time Frame: Baseline, Week 13 (Part 1 and 2)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mcg/kg | Tanezumab 25 mcg/kg | Tanezumab 50 mcg/kg | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 6 | 14
units on a scale | -15.8 (22.60) | -32.7 (25.39) | -23.6 (22.93) | -33.2 (20.10) | -30.6 (27.65) | -24.4 (27.45)
Statistical Analysis 1: Comparison: Tanezumab 10 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = 11.4, 95% CI 2-sided [-5.1 to 27.9], Standard Error of Mean 8.33
Statistical Analysis 2: Comparison: Tanezumab 25 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -8.1, 95% CI 2-sided [-24.4 to 8.2], Standard Error of Mean 8.25
Statistical Analysis 3: Comparison: Tanezumab 50 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = 2.1, 95% CI 2-sided [-14.2 to 18.4], Standard Error of Mean 8.25
Statistical Analysis 4: Comparison: Tanezumab 100 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -8.1, 95% CI 2-sided [-24.3 to 8.0], Standard Error of Mean 8.16
Statistical Analysis 5: Comparison: Tanezumab 200 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -6.4, 95% CI 2-sided [-27.6 to 14.9], Standard Error of Mean 10.75

37. Primary Outcome: Change From Baseline in Visual Analogue Scale (VAS) Score For Index Knee Pain During Walking in the Past 24 Hours at Week 1
Description: VAS assesses participant responses from 0 to 100 (0 = none to 100 = extreme) with 101 point resolution for measuring pain intensity. Higher score indicated greater pain intensity. VAS for index knee pain during walking in the past 24 hours was recorded on the electronic diary.
Time Frame: Baseline, Week 1 (Part 1 and 2)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mcg/kg | Tanezumab 25 mcg/kg | Tanezumab 50 mcg/kg | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 6 | 14
units on a scale
  Baseline | 74.9 (10.11) | 69.4 (10.46) | 72.3 (6.58) | 69.3 (10.45) | 75.5 (7.55) | 69.9 (14.58)
  Change at Week 1 | -18.1 (20.95) | -31.0 (22.33) | -17.7 (20.48) | -26.7 (21.77) | -52.9 (19.71) | -11.0 (11.11)
Statistical Analysis 1: Comparison: Tanezumab 10 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -4.9, 95% CI 2-sided [-21.6 to 11.8], Standard Error of Mean 8.44
Statistical Analysis 2: Comparison: Tanezumab 25 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -19.5, 95% CI 2-sided [-36.1 to -2.9], Standard Error of Mean 8.40
Statistical Analysis 3: Comparison: Tanezumab 50 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -5.2, 95% CI 2-sided [-21.8 to 11.4], Standard Error of Mean 8.40
Statistical Analysis 4: Comparison: Tanezumab 100 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -15.2, 95% CI 2-sided [-31.6 to 1.2], Standard Error of Mean 8.30
Statistical Analysis 5: Comparison: Tanezumab 200 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -40.8, 95% CI 2-sided [-62.6 to -19.0], Standard Error of Mean 11.02

38. Primary Outcome: Change From Baseline in Visual Analogue Scale (VAS) Score For Index Knee Pain During Walking in the Past 24 Hours at Week 2
Description: as for outcome 37
Time Frame: Baseline, Week 2 (Part 1 and 2)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mcg/kg | Tanezumab 25 mcg/kg | Tanezumab 50 mcg/kg | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 6 | 14
units on a scale | -20.7 (19.66) | -30.7 (25.31) | -12.2 (19.49) | -26.7 (19.80) | -32.3 (24.88) | -14.2 (19.12)
Statistical Analysis 1: Comparison: Tanezumab 10 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -4.2, 95% CI 2-sided [-20.9 to 12.5], Standard Error of Mean 8.44
Statistical Analysis 2: Comparison: Tanezumab 25 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -15.9, 95% CI 2-sided [-32.6 to 0.7], Standard Error of Mean 8.40
Statistical Analysis 3: Comparison: Tanezumab 50 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = 3.5, 95% CI 2-sided [-13.2 to 20.1], Standard Error of Mean 8.40
Statistical Analysis 4: Comparison: Tanezumab 100 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -12.0, 95% CI 2-sided [-28.4 to 4.5], Standard Error of Mean 8.30
Statistical Analysis 5: Comparison: Tanezumab 200 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -17.0, 95% CI 2-sided [-38.8 to 4.8], Standard Error of Mean 11.02

39. Primary Outcome: Change From Baseline in Visual Analogue Scale (VAS) Score For Index Knee Pain During Walking in the Past 24 Hours at Week 3
Description: as for outcome 37
Time Frame: Baseline, Week 3 (Part 1 and 2)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mcg/kg | Tanezumab 25 mcg/kg | Tanezumab 50 mcg/kg | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 6 | 14
units on a scale | -24.6 (19.91) | -36.9 (24.37) | -17.3 (22.32) | -29.1 (18.23) | -26.3 (26.71) | -16.9 (22.79)
Statistical Analysis 1: Comparison: Tanezumab 10 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -5.5, 95% CI 2-sided [-22.2 to 11.2], Standard Error of Mean 8.44
Statistical Analysis 2: Comparison: Tanezumab 25 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -19.5, 95% CI 2-sided [-36.1 to -2.9], Standard Error of Mean 8.40
Statistical Analysis 3: Comparison: Tanezumab 50 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = 1.1, 95% CI 2-sided [-15.6 to 17.7], Standard Error of Mean 8.40
Statistical Analysis 4: Comparison: Tanezumab 100 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -11.6, 95% CI 2-sided [-28.0 to 4.8], Standard Error of Mean 8.30
Statistical Analysis 5: Comparison: Tanezumab 200 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -8.3, 95% CI 2-sided [-30.1 to 13.5], Standard Error of Mean 11.02

40. Primary Outcome: Change From Baseline in Visual Analogue Scale (VAS) Score For Index Knee Pain During Walking in the Past 24 Hours at Week 4
Description: as for outcome 37
Time Frame: Baseline, Week 4 (Part 1 and 2)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mcg/kg | Tanezumab 25 mcg/kg | Tanezumab 50 mcg/kg | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 6 | 14
units on a scale | -24.4 (19.88) | -37.8 (26.43) | -22.7 (20.63) | -33.3 (18.10) | -48.8 (19.41) | -18.3 (24.02)
Statistical Analysis 1: Comparison: Tanezumab 10 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -3.9, 95% CI 2-sided [-20.6 to 12.8], Standard Error of Mean 8.44
Statistical Analysis 2: Comparison: Tanezumab 25 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -19.0, 95% CI 2-sided [-35.6 to -2.3], Standard Error of Mean 8.40
Statistical Analysis 3: Comparison: Tanezumab 50 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -2.9, 95% CI 2-sided [-19.6 to 13.7], Standard Error of Mean 8.40
Statistical Analysis 4: Comparison: Tanezumab 100 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -14.5, 95% CI 2-sided [-30.9 to 1.9], Standard Error of Mean 8.30
Statistical Analysis 5: Comparison: Tanezumab 200 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -29.4, 95% CI 2-sided [-51.2 to -7.6], Standard Error of Mean 11.02

41. Primary Outcome: Change From Baseline in Visual Analogue Scale (VAS) Score For Index Knee Pain During Walking in the Past 24 Hours at Week 5
Description: as for outcome 37
Time Frame: Baseline, Week 5 (Part 1 and 2)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mcg/kg | Tanezumab 25 mcg/kg | Tanezumab 50 mcg/kg | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 6 | 14
units on a scale | -21.3 (23.25) | -38.8 (25.14) | -28.4 (24.06) | -35.6 (18.79) | -51.9 (16.04) | -19.5 (25.46)
Statistical Analysis 1: Comparison: Tanezumab 10 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = 0.4, 95% CI 2-sided [-16.3 to 17.1], Standard Error of Mean 8.44
Statistical Analysis 2: Comparison: Tanezumab 25 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -18.8, 95% CI 2-sided [-35.4 to -2.2], Standard Error of Mean 8.40
Statistical Analysis 3: Comparison: Tanezumab 50 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -7.5, 95% CI 2-sided [-24.1 to 9.1], Standard Error of Mean 8.40
Statistical Analysis 4: Comparison: Tanezumab 100 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -15.5, 95% CI 2-sided [-31.9 to 0.9], Standard Error of Mean 8.30
Statistical Analysis 5: Comparison: Tanezumab 200 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -31.3, 95% CI 2-sided [-53.1 to -9.5], Standard Error of Mean 11.02

42. Primary Outcome: Change From Baseline in Visual Analogue Scale (VAS) Score For Index Knee Pain During Walking in the Past 24 Hours at Week 6
Description: as for outcome 37
Time Frame: Baseline, Week 6 (Part 1 and 2)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mcg/kg | Tanezumab 25 mcg/kg | Tanezumab 50 mcg/kg | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 6 | 14
units on a scale | -22.2 (24.42) | -40.3 (25.30) | -28.9 (24.71) | -33.7 (17.08) | -54.7 (15.52) | -19.8 (26.62)
Statistical Analysis 1: Comparison: Tanezumab 10 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -0.2, 95% CI 2-sided [-16.9 to 16.5], Standard Error of Mean 8.44
Statistical Analysis 2: Comparison: Tanezumab 25 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -20.0, 95% CI 2-sided [-36.7 to -3.4], Standard Error of Mean 8.40
Statistical Analysis 3: Comparison: Tanezumab 50 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -7.6, 95% CI 2-sided [-24.2 to 9.0], Standard Error of Mean 8.40
Statistical Analysis 4: Comparison: Tanezumab 100 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -13.4, 95% CI 2-sided [-29.8 to 3.0], Standard Error of Mean 8.30
Statistical Analysis 5: Comparison: Tanezumab 200 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -33.8, 95% CI 2-sided [-55.6 to -12.0], Standard Error of Mean 11.02

43. Primary Outcome: Change From Baseline in Visual Analogue Scale (VAS) Score For Index Knee Pain During Walking in the Past 24 Hours at Week 7
Description: as for outcome 37
Time Frame: Baseline, Week 7 (Part 1 and 2)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mcg/kg | Tanezumab 25 mcg/kg | Tanezumab 50 mcg/kg | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 6 | 14
units on a scale | -18.6 (22.81) | -40.5 (24.92) | -28.2 (24.38) | -35.4 (18.34) | -49.4 (15.06) | -20.1 (27.28)
Statistical Analysis 1: Comparison: Tanezumab 10 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = 3.8, 95% CI 2-sided [-12.9 to 20.4], Standard Error of Mean 8.44
Statistical Analysis 2: Comparison: Tanezumab 25 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -19.9, 95% CI 2-sided [-36.5 to -3.3], Standard Error of Mean 8.40
Statistical Analysis 3: Comparison: Tanezumab 50 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -6.7, 95% CI 2-sided [-23.3 to 10.0], Standard Error of Mean 8.40
Statistical Analysis 4: Comparison: Tanezumab 100 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -14.8, 95% CI 2-sided [-31.2 to 1.6], Standard Error of Mean 8.30
Statistical Analysis 5: Comparison: Tanezumab 200 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -28.2, 95% CI 2-sided [-50.0 to -6.4], Standard Error of Mean 11.02

44. Primary Outcome: Change From Baseline in Visual Analogue Scale (VAS) Score For Index Knee Pain During Walking in the Past 24 Hours at Week 8
Description: as for outcome 37
Time Frame: Baseline, Week 8 (Part 1 and 2)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mcg/kg | Tanezumab 25 mcg/kg | Tanezumab 50 mcg/kg | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 6 | 14
units on a scale | -17.5 (23.15) | -40.9 (25.00) | -27.3 (23.85) | -36.6 (19.21) | -52.1 (18.37) | -22.5 (26.93)
Statistical Analysis 1: Comparison: Tanezumab 10 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = 7.3, 95% CI 2-sided [-9.4 to 24.0], Standard Error of Mean 8.44
Statistical Analysis 2: Comparison: Tanezumab 25 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -17.8, 95% CI 2-sided [-34.4 to -1.2], Standard Error of Mean 8.40
Statistical Analysis 3: Comparison: Tanezumab 50 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -3.4, 95% CI 2-sided [-20.0 to 13.2], Standard Error of Mean 8.40
Statistical Analysis 4: Comparison: Tanezumab 100 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -13.5, 95% CI 2-sided [-29.9 to 2.9], Standard Error of Mean 8.30
Statistical Analysis 5: Comparison: Tanezumab 200 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -28.5, 95% CI 2-sided [-50.3 to -6.7], Standard Error of Mean 11.02

45. Primary Outcome: Change From Baseline in Visual Analogue Scale (VAS) Score For Index Knee Pain During Walking in the Past 24 Hours at Week 9
Description: as for outcome 37
Time Frame: Baseline, Week 9 (Part 1 and 2)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mcg/kg | Tanezumab 25 mcg/kg | Tanezumab 50 mcg/kg | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 6 | 14
units on a scale | -16.4 (22.80) | -41.8 (27.37) | -25.9 (21.91) | -35.6 (20.43) | -50.7 (14.75) | -26.5 (27.46)
Statistical Analysis 1: Comparison: Tanezumab 10 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = 12.4, 95% CI 2-sided [-4.3 to 29.1], Standard Error of Mean 8.44
Statistical Analysis 2: Comparison: Tanezumab 25 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -14.8, 95% CI 2-sided [-31.4 to 1.9], Standard Error of Mean 8.40
Statistical Analysis 3: Comparison: Tanezumab 50 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = 2.0, 95% CI 2-sided [-14.6 to 18.6], Standard Error of Mean 8.40
Statistical Analysis 4: Comparison: Tanezumab 100 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -8.6, 95% CI 2-sided [-25.0 to 7.8], Standard Error of Mean 8.30
Statistical Analysis 5: Comparison: Tanezumab 200 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -23.1, 95% CI 2-sided [-44.9 to -1.3], Standard Error of Mean 11.02

46. Primary Outcome: Change From Baseline in Visual Analogue Scale (VAS) Score For Index Knee Pain During Walking in the Past 24 Hours at Week 10
Description: as for outcome 37
Time Frame: Baseline, Week 10 (Part 1 and 2)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mcg/kg | Tanezumab 25 mcg/kg | Tanezumab 50 mcg/kg | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 6 | 14
units on a scale | -15.5 (20.29) | -40.8 (29.14) | -23.2 (21.04) | -32.1 (20.85) | -44.9 (18.13) | -24.8 (27.21)
Statistical Analysis 1: Comparison: Tanezumab 10 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = 11.6, 95% CI 2-sided [-5.1 to 28.3], Standard Error of Mean 8.44
Statistical Analysis 2: Comparison: Tanezumab 25 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -15.5, 95% CI 2-sided [-32.1 to 1.1], Standard Error of Mean 8.40
Statistical Analysis 3: Comparison: Tanezumab 50 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = 3.1, 95% CI 2-sided [-13.5 to 19.7], Standard Error of Mean 8.40
Statistical Analysis 4: Comparison: Tanezumab 100 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -6.7, 95% CI 2-sided [-23.1 to 9.7], Standard Error of Mean 8.30
Statistical Analysis 5: Comparison: Tanezumab 200 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -18.9, 95% CI 2-sided [-40.7 to 2.9], Standard Error of Mean 11.02

47. Primary Outcome: Change From Baseline in Visual Analogue Scale (VAS) Score For Index Knee Pain During Walking in the Past 24 Hours at Week 11
Description: as for outcome 37
Time Frame: Baseline, Week 11 (Part 1 and 2)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mcg/kg | Tanezumab 25 mcg/kg | Tanezumab 50 mcg/kg | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 6 | 14
units on a scale | -15.1 (16.52) | -36.8 (25.95) | -23.1 (20.80) | -33.1 (19.01) | -44.8 (21.86) | -25.1 (26.19)
Statistical Analysis 1: Comparison: Tanezumab 10 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = 12.3, 95% CI 2-sided [-4.4 to 29.0], Standard Error of Mean 8.44
Statistical Analysis 2: Comparison: Tanezumab 25 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -11.2, 95% CI 2-sided [-27.8 to 5.4], Standard Error of Mean 8.40
Statistical Analysis 3: Comparison: Tanezumab 50 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = 3.5, 95% CI 2-sided [-13.2 to 20.1], Standard Error of Mean 8.40
Statistical Analysis 4: Comparison: Tanezumab 100 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -7.5, 95% CI 2-sided [-23.9 to 9.0], Standard Error of Mean 8.30
Statistical Analysis 5: Comparison: Tanezumab 200 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -18.6, 95% CI 2-sided [-40.4 to 3.2], Standard Error of Mean 11.02

48. Primary Outcome: Change From Baseline in Visual Analogue Scale (VAS) Score For Index Knee Pain During Walking in the Past 24 Hours at Week 12
Description: as for outcome 37
Time Frame: Baseline, Week 12 (Part 1 and 2)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mcg/kg | Tanezumab 25 mcg/kg | Tanezumab 50 mcg/kg | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 6 | 14
units on a scale | -15.0 (16.67) | -34.1 (24.63) | -23.5 (20.35) | -31.6 (19.93) | -45.4 (24.54) | -23.9 (27.70)
Statistical Analysis 1: Comparison: Tanezumab 10 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = 11.2, 95% CI 2-sided [-5.5 to 27.9], Standard Error of Mean 8.44
Statistical Analysis 2: Comparison: Tanezumab 25 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -9.6, 95% CI 2-sided [-26.3 to 7.0], Standard Error of Mean 8.40
Statistical Analysis 3: Comparison: Tanezumab 50 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = 1.9, 95% CI 2-sided [-14.7 to 18.5], Standard Error of Mean 8.40
Statistical Analysis 4: Comparison: Tanezumab 100 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -7.2, 95% CI 2-sided [-23.6 to 9.2], Standard Error of Mean 8.30
Statistical Analysis 5: Comparison: Tanezumab 200 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -20.4, 95% CI 2-sided [-42.2 to 1.4], Standard Error of Mean 11.02

49. Primary Outcome: Change From Baseline in Visual Analogue Scale (VAS) Score For Index Knee Pain During Walking in the Past 24 Hours at Week 13
Description: as for outcome 37
Time Frame: Baseline, Week 13 (Part 1 and 2)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mcg/kg | Tanezumab 25 mcg/kg | Tanezumab 50 mcg/kg | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 6 | 14
units on a scale | -13.1 (21.25) | -31.5 (25.99) | -20.7 (19.36) | -32.7 (21.74) | -35.3 (34.29) | -24.3 (29.09)
Statistical Analysis 1: Comparison: Tanezumab 10 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = 13.5, 95% CI 2-sided [-3.2 to 30.2], Standard Error of Mean 8.44
Statistical Analysis 2: Comparison: Tanezumab 25 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -6.7, 95% CI 2-sided [-23.3 to 9.9], Standard Error of Mean 8.40
Statistical Analysis 3: Comparison: Tanezumab 50 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = 5.1, 95% CI 2-sided [-11.5 to 21.7], Standard Error of Mean 8.40
Statistical Analysis 4: Comparison: Tanezumab 100 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -7.6, 95% CI 2-sided [-24.1 to 8.8], Standard Error of Mean 8.31
Statistical Analysis 5: Comparison: Tanezumab 200 mcg/kg vs Placebo; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -9.8, 95% CI 2-sided [-31.6 to 12.0], Standard Error of Mean 11.02

50. Primary Outcome: Change From Baseline in Western Ontario and McMaster Universities Osteoarthritis Version 3.1 (WOMAC 3.1) Subscales Scores at Week 1
Description: WOMAC 3.1: participant assessed questionnaire consists of 24 questions divided into 3 domains; pain (5 questions), stiffness (2 questions), function (17 questions). Functional domain provided information of ability to perform activities of daily living. The participant performed test directly on electronic diary, using validated electronic VAS ranging from 0 to 100 (0 = none to 100 = extreme). Each domain scored by averaging VAS scores of component questions. Total subscale score for each of the 3 domains range from: 0 to 100, lower score indicated better daily living.
Time Frame: Baseline, Week 1 (Part 1 and 2)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mcg/kg | Tanezumab 25 mcg/kg | Tanezumab 50 mcg/kg | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 6 | 14
units on a scale
  Baseline: Pain | 61.3 (16.33) | 61.0 (16.29) | 65.2 (11.07) | 58.0 (13.04) | 59.2 (16.81) | 54.1 (17.70)
  Baseline: Physical Function | 55.8 (19.88) | 56.0 (13.22) | 67.8 (8.94) | 60.5 (17.94) | 57.8 (18.26) | 53.4 (14.85)
  Baseline: Stiffness | 50.7 (18.78) | 50.7 (20.86) | 69.5 (11.86) | 56.2 (23.86) | 55.3 (22.24) | 54.2 (21.89)
  Change at Week 1: Pain | -19.5 (24.89) | -30.6 (23.79) | -16.2 (22.63) | -24.6 (17.94) | -37.1 (20.94) | -6.4 (11.18)
  Change at Week 1: Physical Function | -13.9 (29.69) | -26.6 (22.15) | -19.0 (20.68) | -27.3 (19.45) | -35.2 (29.04) | -10.6 (14.69)
  Change at Week 1: Stiffness | -17.5 (33.85) | -27.9 (30.09) | -21.9 (29.86) | -24.2 (23.29) | -30.7 (28.30) | -4.4 (19.93)
Statistical Analysis 1: Comparison: Tanezumab 10 mcg/kg vs Placebo; Change at Week 1, Pain: Mixed Model for Repeated Measures analyses included fixed effects of treatment, week, treatment by week, part, and baseline values; Test type: Superiority or Other; Least Square Mean Difference = -9.2, 95% CI 2-sided [-24.7 to 6.4], Standard Error of Mean 7.86
Statistical Analysis 2: Comparison: Tanezumab 25 mcg/kg vs Placebo; [analysis description as in outcome 50, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -20.4, 95% CI 2-sided [-36.0 to -4.9], Standard Error of Mean 7.86
Statistical Analysis 3: Comparison: Tanezumab 50 mcg/kg vs Placebo; [analysis description as in outcome 50, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -4.2, 95% CI 2-sided [-19.9 to 11.4], Standard Error of Mean 7.92
Statistical Analysis 4: Comparison: Tanezumab 100 mcg/kg vs Placebo; [analysis description as in outcome 50, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -15.7, 95% CI 2-sided [-30.9 to -0.4], Standard Error of Mean 7.73
Statistical Analysis 5: Comparison: Tanezumab 200 mcg/kg vs Placebo; [analysis description as in outcome 50, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -29.1, 95% CI 2-sided [-49.4 to -8.9], Standard Error of Mean 10.25
Statistical Analysis 6: Comparison: Tanezumab 10 mcg/kg vs Placebo; Change at Week 1, Physical Functions: Mixed Model for Repeated Measures analyses included fixed effects of treatment, week, treatment by week, part, and baseline values; Test type: Superiority or Other; Least Square Mean Difference = -1.3, 95% CI 2-sided [-16.9 to 14.3], Standard Error of Mean 7.89
Statistical Analysis 7: Comparison: Tanezumab 25 mcg/kg vs Placebo; [analysis description as in outcome 50, analysis 6]; Test type: Superiority or Other; Least Square Mean Difference = -13.9, 95% CI 2-sided [-29.5 to 1.7], Standard Error of Mean 7.89
Statistical Analysis 8: Comparison: Tanezumab 50 mcg/kg vs Placebo; [analysis description as in outcome 50, analysis 6]; Test type: Superiority or Other; Least Square Mean Difference = 0.6, 95% CI 2-sided [-15.4 to 16.5], Standard Error of Mean 8.06
Statistical Analysis 9: Comparison: Tanezumab 100 mcg/kg vs Placebo; [analysis description as in outcome 50, analysis 6]; Test type: Superiority or Other; Least Square Mean Difference = -11.8, 95% CI 2-sided [-27.3 to 3.7], Standard Error of Mean 7.83
Statistical Analysis 10: Comparison: Tanezumab 200 mcg/kg vs Placebo; [analysis description as in outcome 50, analysis 6]; Test type: Superiority or Other; Least Square Mean Difference = -22.7, 95% CI 2-sided [-43.1 to -2.4], Standard Error of Mean 10.30
Statistical Analysis 11: Comparison: Tanezumab 10 mcg/kg vs Placebo; Change at Week 1, Stiffness: Mixed Model for Repeated Measures analyses included fixed effects of treatment, week, treatment by week, part, and baseline values; Test type: Superiority or Other; Least Square Mean Difference = -16.7, 95% CI 2-sided [-33.2 to -0.3], Standard Error of Mean 8.34
Statistical Analysis 12: Comparison: Tanezumab 25 mcg/kg vs Placebo; [analysis description as in outcome 50, analysis 11]; Test type: Superiority or Other; Least Square Mean Difference = -27.2, 95% CI 2-sided [-43.7 to -10.8], Standard Error of Mean 8.34
Statistical Analysis 13: Comparison: Tanezumab 50 mcg/kg vs Placebo; [analysis description as in outcome 50, analysis 11]; Test type: Superiority or Other; Least Square Mean Difference = -6.8, 95% CI 2-sided [-23.4 to 9.9], Standard Error of Mean 8.45
Statistical Analysis 14: Comparison: Tanezumab 100 mcg/kg vs Placebo; [analysis description as in outcome 50, analysis 11]; Test type: Superiority or Other; Least Square Mean Difference = -19.4, 95% CI 2-sided [-35.6 to -3.2], Standard Error of Mean 8.22
Statistical Analysis 15: Comparison: Tanezumab 200 mcg/kg vs Placebo; [analysis description as in outcome 50, analysis 11]; Test type: Superiority or Other; Least Square Mean Difference = -24.4, 95% CI 2-sided [-45.8 to -2.9], Standard Error of Mean 10.86

51. Primary Outcome: Change From Baseline in WOMAC 3.1 Subscales Scores at Week 2
Description: as for outcome 50
Time Frame: Baseline, Week 2 (Part 1 and 2)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mcg/kg | Tanezumab 25 mcg/kg | Tanezumab 50 mcg/kg | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 6 | 14
units on a scale
  Change at Week 2: Pain | -16.8 (19.88) | -28.5 (25.69) | -3.1 (25.93) | -20.3 (18.51) | -14.5 (18.74) | -10.0 (15.90)
  Change at Week 2: Physical Function | -12.8 (25.96) | -23.5 (23.65) | -7.9 (20.46) | -22.8 (18.16) | -18.2 (23.96) | -11.4 (18.53)
  Change at Week 2: Stiffness | -15.4 (29.13) | -24.3 (25.23) | -8.8 (25.35) | -21.3 (19.68) | -20.1 (35.94) | -14.2 (22.34)
Statistical Analysis 1: Comparison: Tanezumab 10 mcg/kg vs Placebo; Change at Week 2, Pain: Mixed Model for Repeated Measures analyses included fixed effects of treatment, week, treatment by week, part, and baseline values; Test type: Superiority or Other; Least Square Mean Difference = -2.9, 95% CI 2-sided [-18.5 to 12.6], Standard Error of Mean 7.86
Statistical Analysis 2: Comparison: Tanezumab 25 mcg/kg vs Placebo; [analysis description as in outcome 51, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -14.7, 95% CI 2-sided [-30.3 to 0.8], Standard Error of Mean 7.86
Statistical Analysis 3: Comparison: Tanezumab 50 mcg/kg vs Placebo; [analysis description as in outcome 51, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = 12.4, 95% CI 2-sided [-3.2 to 28.1], Standard Error of Mean 7.92
Statistical Analysis 4: Comparison: Tanezumab 100 mcg/kg vs Placebo; [analysis description as in outcome 51, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -7.8, 95% CI 2-sided [-23.1 to 7.4], Standard Error of Mean 7.73
Statistical Analysis 5: Comparison: Tanezumab 200 mcg/kg vs Placebo; [analysis description as in outcome 51, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -3.0, 95% CI 2-sided [-23.3 to 17.2], Standard Error of Mean 10.25
Statistical Analysis 6: Comparison: Tanezumab 10 mcg/kg vs Placebo; Change at Week 2, Physical functions: Mixed Model for Repeated Measures analyses included fixed effects of treatment, week, treatment by week, part, and baseline values; Test type: Superiority or Other; Least Square Mean Difference = 0.7, 95% CI 2-sided [-14.9 to 16.3], Standard Error of Mean 7.89
Statistical Analysis 7: Comparison: Tanezumab 25 mcg/kg vs Placebo; [analysis description as in outcome 51, analysis 6]; Test type: Superiority or Other; Least Square Mean Difference = -9.9, 95% CI 2-sided [-25.5 to 5.7], Standard Error of Mean 7.89
Statistical Analysis 8: Comparison: Tanezumab 50 mcg/kg vs Placebo; [analysis description as in outcome 51, analysis 6]; Test type: Superiority or Other; Least Square Mean Difference = 12.5, 95% CI 2-sided [-3.4 to 28.5], Standard Error of Mean 8.06
Statistical Analysis 9: Comparison: Tanezumab 100 mcg/kg vs Placebo; [analysis description as in outcome 51, analysis 6]; Test type: Superiority or Other; Least Square Mean Difference = -6.5, 95% CI 2-sided [-21.9 to 9.0], Standard Error of Mean 7.83
Statistical Analysis 10: Comparison: Tanezumab 200 mcg/kg vs Placebo; [analysis description as in outcome 51, analysis 6]; Test type: Superiority or Other; Least Square Mean Difference = -4.9, 95% CI 2-sided [-25.2 to 15.5], Standard Error of Mean 10.30
Statistical Analysis 11: Comparison: Tanezumab 10 mcg/kg vs Placebo; Change at Week 2, Stiffness: Mixed Model for Repeated Measures analyses included fixed effects of treatment, week, treatment by week, part, and baseline values; Test type: Superiority or Other; Least Square Mean Difference = -5.0, 95% CI 2-sided [-21.4 to 11.5], Standard Error of Mean 8.34
Statistical Analysis 12: Comparison: Tanezumab 25 mcg/kg vs Placebo; [analysis description as in outcome 51, analysis 11]; Test type: Superiority or Other; Least Square Mean Difference = -13.8, 95% CI 2-sided [-30.3 to 2.7], Standard Error of Mean 8.34
Statistical Analysis 13: Comparison: Tanezumab 50 mcg/kg vs Placebo; [analysis description as in outcome 51, analysis 11]; Test type: Superiority or Other; Least Square Mean Difference = 16.1, 95% CI 2-sided [-0.6 to 32.7], Standard Error of Mean 8.45
Statistical Analysis 14: Comparison: Tanezumab 100 mcg/kg vs Placebo; [analysis description as in outcome 51, analysis 11]; Test type: Superiority or Other; Least Square Mean Difference = -6.7, 95% CI 2-sided [-22.9 to 9.5], Standard Error of Mean 8.22
Statistical Analysis 15: Comparison: Tanezumab 200 mcg/kg vs Placebo; [analysis description as in outcome 51, analysis 11]; Test type: Superiority or Other; Least Square Mean Difference = -4.0, 95% CI 2-sided [-25.5 to 17.4], Standard Error of Mean 10.86

52. Primary Outcome: Change From Baseline in WOMAC 3.1 Subscales Scores at Week 4
Description: as for outcome 50
Time Frame: Baseline, Week 4 (Part 1 and 2)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mcg/kg | Tanezumab 25 mcg/kg | Tanezumab 50 mcg/kg | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 6 | 14
units on a scale
  Change at Week 4: Pain | -23.7 (22.84) | -35.1 (24.91) | -27.6 (25.39) | -30.4 (16.35) | -41.9 (15.65) | -12.5 (19.83)
  Change at Week 4: Physical Function | -19.3 (28.10) | -30.8 (24.23) | -29.0 (24.93) | -33.3 (19.20) | -41.0 (21.33) | -11.6 (24.67)
  Change at Week 4: Stiffness | -19.6 (32.36) | -30.2 (28.81) | -30.3 (29.00) | -29.3 (21.58) | -39.1 (31.46) | -14.3 (26.04)
Statistical Analysis 1: Comparison: Tanezumab 10 mcg/kg vs Placebo; Change at Week 4, Pain: Mixed Model for Repeated Measures analyses included fixed effects of treatment, week, treatment by week, part, and baseline values; Test type: Superiority or Other; Least Square Mean Difference = -7.3, 95% CI 2-sided [-22.9 to 8.2], Standard Error of Mean 7.86
Statistical Analysis 2: Comparison: Tanezumab 25 mcg/kg vs Placebo; [analysis description as in outcome 52, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -18.9, 95% CI 2-sided [-34.4 to -3.3], Standard Error of Mean 7.86
Statistical Analysis 3: Comparison: Tanezumab 50 mcg/kg vs Placebo; [analysis description as in outcome 52, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -9.6, 95% CI 2-sided [-25.2 to 6.1], Standard Error of Mean 7.92
Statistical Analysis 4: Comparison: Tanezumab 100 mcg/kg vs Placebo; [analysis description as in outcome 52, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -15.5, 95% CI 2-sided [-30.8 to -0.2], Standard Error of Mean 7.73
Statistical Analysis 5: Comparison: Tanezumab 200 mcg/kg vs Placebo; [analysis description as in outcome 52, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -27.9, 95% CI 2-sided [-48.1 to -7.6], Standard Error of Mean 10.25
Statistical Analysis 6: Comparison: Tanezumab 10 mcg/kg vs Placebo; Change at Week 4, Physical Functions: Mixed Model for Repeated Measures analyses included fixed effects of treatment, week, treatment by week, part, and baseline values; Test type: Superiority or Other; Least Square Mean Difference = -5.7, 95% CI 2-sided [-21.3 to 9.9], Standard Error of Mean 7.89
Statistical Analysis 7: Comparison: Tanezumab 25 mcg/kg vs Placebo; [analysis description as in outcome 52, analysis 6]; Test type: Superiority or Other; Least Square Mean Difference = -17.0, 95% CI 2-sided [-32.6 to -1.4], Standard Error of Mean 7.89
Statistical Analysis 8: Comparison: Tanezumab 50 mcg/kg vs Placebo; [analysis description as in outcome 52, analysis 6]; Test type: Superiority or Other; Least Square Mean Difference = -8.4, 95% CI 2-sided [-24.3 to 7.5], Standard Error of Mean 8.06
Statistical Analysis 9: Comparison: Tanezumab 100 mcg/kg vs Placebo; [analysis description as in outcome 52, analysis 6]; Test type: Superiority or Other; Least Square Mean Difference = -16.8, 95% CI 2-sided [-32.2 to -1.3], Standard Error of Mean 7.83
Statistical Analysis 10: Comparison: Tanezumab 200 mcg/kg vs Placebo; [analysis description as in outcome 52, analysis 6]; Test type: Superiority or Other; Least Square Mean Difference = -27.5, 95% CI 2-sided [-47.8 to -7.1], Standard Error of Mean 10.30
Statistical Analysis 11: Comparison: Tanezumab 10 mcg/kg vs Placebo; Change at Week 4, Stiffness: Mixed Model for Repeated Measures analyses included fixed effects of treatment, week, treatment by week, part, and baseline values; Test type: Superiority or Other; Least Square Mean Difference = -9.0, 95% CI 2-sided [-25.5 to 7.4], Standard Error of Mean 8.34
Statistical Analysis 12: Comparison: Tanezumab 25 mcg/kg vs Placebo; [analysis description as in outcome 52, analysis 11]; Test type: Superiority or Other; Least Square Mean Difference = -19.7, 95% CI 2-sided [-36.1 to -3.2], Standard Error of Mean 8.34
Statistical Analysis 13: Comparison: Tanezumab 50 mcg/kg vs Placebo; [analysis description as in outcome 52, analysis 11]; Test type: Superiority or Other; Least Square Mean Difference = -5.4, 95% CI 2-sided [-22.1 to 11.3], Standard Error of Mean 8.45
Statistical Analysis 14: Comparison: Tanezumab 100 mcg/kg vs Placebo; [analysis description as in outcome 52, analysis 11]; Test type: Superiority or Other; Least Square Mean Difference = -14.7, 95% CI 2-sided [-30.9 to 1.6], Standard Error of Mean 8.22
Statistical Analysis 15: Comparison: Tanezumab 200 mcg/kg vs Placebo; [analysis description as in outcome 52, analysis 11]; Test type: Superiority or Other; Least Square Mean Difference = -23.0, 95% CI 2-sided [-44.4 to -1.5], Standard Error of Mean 10.86

53. Primary Outcome: Change From Baseline in WOMAC 3.1 Subscales Scores at Week 8
Description: WOMAC 3.1: participant assessed questionnaire consists of 24 questions divided into 3 domains; pain (5 questions), stiffness (2 questions), function (17 questions). Functional domain provided information of ability to perform activities of daily living. The participant performed test directly on electronic diary, using validated electronic VAS ranging from 0 to 100 (0=none to 100= extreme). Each domain scored by averaging VAS scores of component questions. Total subscale score for each of the 3 domains range from: 0 to 100, lower score indicated better daily living.
Time Frame: Baseline, Week 8 (Part 1 and 2)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mcg/kg | Tanezumab 25 mcg/kg | Tanezumab 50 mcg/kg | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 6 | 14
units on a scale
  Change at Week 8: Pain | -20.7 (20.64) | -35.3 (25.28) | -27.4 (26.62) | -32.1 (16.07) | -40.6 (21.08) | -20.1 (19.11)
  Change at Week 8: Physical Function | -16.3 (18.65) | -29.9 (26.89) | -29.4 (23.71) | -33.3 (19.49) | -39.0 (21.10) | -19.3 (19.81)
  Change at Week 8: Stiffness | -16.8 (24.56) | -35.1 (25.39) | -32.2 (29.58) | -30.0 (19.41) | -31.1 (27.18) | -18.7 (23.16)
Statistical Analysis 1: Comparison: Tanezumab 10 mcg/kg vs Placebo; Change at Week 8, Pain: Mixed Model for Repeated Measures analyses included fixed effects of treatment, week, treatment by week, part, and baseline values; Test type: Superiority or Other; Least Square Mean Difference = 3.3, 95% CI 2-sided [-12.2 to 18.8], Standard Error of Mean 7.86
Statistical Analysis 2: Comparison: Tanezumab 25 mcg/kg vs Placebo; [analysis description as in outcome 53, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -11.4, 95% CI 2-sided [-27.0 to 4.1], Standard Error of Mean 7.86
Statistical Analysis 3: Comparison: Tanezumab 50 mcg/kg vs Placebo; [analysis description as in outcome 53, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -1.7, 95% CI 2-sided [-17.4 to 13.9], Standard Error of Mean 7.92
Statistical Analysis 4: Comparison: Tanezumab 100 mcg/kg vs Placebo; [analysis description as in outcome 53, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -9.5, 95% CI 2-sided [-24.8 to 5.8], Standard Error of Mean 7.73
Statistical Analysis 5: Comparison: Tanezumab 200 mcg/kg vs Placebo; [analysis description as in outcome 53, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -19.0, 95% CI 2-sided [-39.2 to 1.3], Standard Error of Mean 10.25
Statistical Analysis 6: Comparison: Tanezumab 10 mcg/kg vs Placebo; Change at Week 8, Physical functions: Mixed Model for Repeated Measures analyses included fixed effects of treatment, week, treatment by week, part, and baseline values; Test type: Superiority or Other; Least Square Mean Difference = 5.0, 95% CI 2-sided [-10.6 to 20.6], Standard Error of Mean 7.89
Statistical Analysis 7: Comparison: Tanezumab 25 mcg/kg vs Placebo; [analysis description as in outcome 53, analysis 6]; Test type: Superiority or Other; Least Square Mean Difference = -8.4, 95% CI 2-sided [-24.0 to 7.1], Standard Error of Mean 7.89
Statistical Analysis 8: Comparison: Tanezumab 50 mcg/kg vs Placebo; [analysis description as in outcome 53, analysis 6]; Test type: Superiority or Other; Least Square Mean Difference = -1.2, 95% CI 2-sided [-17.1 to 14.8], Standard Error of Mean 8.06
Statistical Analysis 9: Comparison: Tanezumab 100 mcg/kg vs Placebo; [analysis description as in outcome 53, analysis 6]; Test type: Superiority or Other; Least Square Mean Difference = -9.2, 95% CI 2-sided [-24.6 to 6.3], Standard Error of Mean 7.83
Statistical Analysis 10: Comparison: Tanezumab 200 mcg/kg vs Placebo; [analysis description as in outcome 53, analysis 6]; Test type: Superiority or Other; Least Square Mean Difference = -17.8, 95% CI 2-sided [-38.2 to 2.5], Standard Error of Mean 10.30
Statistical Analysis 11: Comparison: Tanezumab 10 mcg/kg vs Placebo; Change at Week 8, Stiffness: Mixed Model for Repeated Measures analyses included fixed effects of treatment, week, treatment by week, part, and baseline values; Test type: Superiority or Other; Least Square Mean Difference = -1.8, 95% CI 2-sided [-18.3 to 14.6], Standard Error of Mean 8.34
Statistical Analysis 12: Comparison: Tanezumab 25 mcg/kg vs Placebo; [analysis description as in outcome 53, analysis 11]; Test type: Superiority or Other; Least Square Mean Difference = -20.1, 95% CI 2-sided [-36.5 to -3.6], Standard Error of Mean 8.34
Statistical Analysis 13: Comparison: Tanezumab 50 mcg/kg vs Placebo; [analysis description as in outcome 53, analysis 11]; Test type: Superiority or Other; Least Square Mean Difference = -2.8, 95% CI 2-sided [-19.5 to 13.9], Standard Error of Mean 8.45
Statistical Analysis 14: Comparison: Tanezumab 100 mcg/kg vs Placebo; [analysis description as in outcome 53, analysis 11]; Test type: Superiority or Other; Least Square Mean Difference = -10.9, 95% CI 2-sided [-27.1 to 5.4], Standard Error of Mean 8.22
Statistical Analysis 15: Comparison: Tanezumab 200 mcg/kg vs Placebo; [analysis description as in outcome 53, analysis 11]; Test type: Superiority or Other; Least Square Mean Difference = -10.5, 95% CI 2-sided [-32.0 to 10.9], Standard Error of Mean 10.86

54. Primary Outcome: Change From Baseline in WOMAC 3.1 Subscales Scores at Week 13
Description: as for outcome 50
Time Frame: Baseline, Week 13 (Part 1 and 2)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 10 mcg/kg | Tanezumab 25 mcg/kg | Tanezumab 50 mcg/kg | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg | Placebo
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 6 | 14
units on a scale
  Change at Week 13: Pain | -8.8 (22.81) | -27.1 (24.64) | -18.2 (21.92) | -28.2 (17.77) | -28.9 (28.82) | -17.9 (25.91)
  Change at Week 13: Physical Function | -4.3 (24.86) | -22.2 (24.70) | -18.6 (19.10) | -31.7 (18.37) | -26.8 (29.62) | -16.5 (25.99)
  Change at Week 13: Stiffness | -7.9 (33.04) | -20.8 (26.16) | -17.0 (21.03) | -27.9 (20.73) | -21.4 (33.51) | -18.6 (28.16)
Statistical Analysis 1: Comparison: Tanezumab 10 mcg/kg vs Placebo; Change at Week 13, Pain: Mixed Model for Repeated Measures analyses included fixed effects of treatment, week, treatment by week, part, and baseline values; Test type: Superiority or Other; Least Square Mean Difference = 13.0, 95% CI 2-sided [-2.5 to 28.6], Standard Error of Mean 7.86
Statistical Analysis 2: Comparison: Tanezumab 25 mcg/kg vs Placebo; [analysis description as in outcome 54, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -5.5, 95% CI 2-sided [-21.0 to 10.0], Standard Error of Mean 7.86
Statistical Analysis 3: Comparison: Tanezumab 50 mcg/kg vs Placebo; [analysis description as in outcome 54, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = 5.3, 95% CI 2-sided [-10.4 to 20.9], Standard Error of Mean 7.92
Statistical Analysis 4: Comparison: Tanezumab 100 mcg/kg vs Placebo; [analysis description as in outcome 54, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -7.8, 95% CI 2-sided [-23.1 to 7.5], Standard Error of Mean 7.73
Statistical Analysis 5: Comparison: Tanezumab 200 mcg/kg vs Placebo; [analysis description as in outcome 54, analysis 1]; Test type: Superiority or Other; Least Square Mean Difference = -9.5, 95% CI 2-sided [-29.7 to 10.8], Standard Error of Mean 10.25
Statistical Analysis 6: Comparison: Tanezumab 10 mcg/kg vs Placebo; Change at Week 13, Physical Functions: Mixed Model for Repeated Measures analyses included fixed effects of treatment, week, treatment by week, part, and baseline values; Test type: Superiority or Other; Least Square Mean Difference = 14.3, 95% CI 2-sided [-1.3 to 29.8], Standard Error of Mean 7.89
Statistical Analysis 7: Comparison: Tanezumab 25 mcg/kg vs Placebo; [analysis description as in outcome 54, analysis 6]; Test type: Superiority or Other; Least Square Mean Difference = -3.6, 95% CI 2-sided [-19.2 to 12.0], Standard Error of Mean 7.89
Statistical Analysis 8: Comparison: Tanezumab 50 mcg/kg vs Placebo; [analysis description as in outcome 54, analysis 6]; Test type: Superiority or Other; Least Square Mean Difference = 6.8, 95% CI 2-sided [-9.1 to 22.8], Standard Error of Mean 8.06
Statistical Analysis 9: Comparison: Tanezumab 100 mcg/kg vs Placebo; [analysis description as in outcome 54, analysis 6]; Test type: Superiority or Other; Least Square Mean Difference = -10.3, 95% CI 2-sided [-25.8 to 5.1], Standard Error of Mean 7.83
Statistical Analysis 10: Comparison: Tanezumab 200 mcg/kg vs Placebo; [analysis description as in outcome 54, analysis 6]; Test type: Superiority or Other; Least Square Mean Difference = -8.4, 95% CI 2-sided [-28.8 to 12.0], Standard Error of Mean 10.30
Statistical Analysis 11: Comparison: Tanezumab 10 mcg/kg vs Placebo; Change at Week 13, Stiffness: Mixed Model for Repeated Measures analyses included fixed effects of treatment, week, treatment by week, part, and baseline values; Test type: Superiority or Other; Least Square Mean Difference = 7.0, 95% CI 2-sided [-9.5 to 23.4], Standard Error of Mean 8.34
Statistical Analysis 12: Comparison: Tanezumab 25 mcg/kg vs Placebo; [analysis description as in outcome 54, analysis 11]; Test type: Superiority or Other; Least Square Mean Difference = -5.9, 95% CI 2-sided [-22.4 to 10.6], Standard Error of Mean 8.34
Statistical Analysis 13: Comparison: Tanezumab 50 mcg/kg vs Placebo; [analysis description as in outcome 54, analysis 11]; Test type: Superiority or Other; Least Square Mean Difference = 12.2, 95% CI 2-sided [-4.5 to 28.9], Standard Error of Mean 8.45
Statistical Analysis 14: Comparison: Tanezumab 100 mcg/kg vs Placebo; [analysis description as in outcome 54, analysis 11]; Test type: Superiority or Other; Least Square Mean Difference = -9.0, 95% CI 2-sided [-25.2 to 7.2], Standard Error of Mean 8.22
Statistical Analysis 15: Comparison: Tanezumab 200 mcg/kg vs Placebo; [analysis description as in outcome 54, analysis 11]; Test type: Superiority or Other; Least Square Mean Difference = -1.0, 95% CI 2-sided [-22.4 to 20.5], Standard Error of Mean 10.86

55. Primary Outcome: Change From Baseline in WOMAC 3.1 Subscales Scores at Week 17
Description: as for outcome 50
Time Frame: Baseline, Week 17 (Part 1 and 2)
Population: FAS. Here, 'overall number of participants analyzed' signifies those who were evaluable for this measure. Week 17: analysis was performed only for treatment arms Tanezumab 100 mcg/kg, 200 mcg/kg and Placebo as per analysis plan. It was planned to report combined data for Part 1 and 2.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg | Placebo
Number analyzed (Participants) | 16 | 6 | 14
units on a scale
  Change at Week 17: Pain | -26.6 (20.14) | -32.3 (18.58) | -41.7 (22.45)
  Change at Week 17: Physical Function | -30.1 (20.99) | -30.1 (24.69) | -36.8 (23.41)
  Change at Week 17: Stiffness | -21.7 (17.50) | -20.3 (27.72) | -43.3 (20.11)

56. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) - Part 1
Time Frame: Part 1: Pre-dose, Day 1 (10 minutes, 0.5, 1, 4, 12 hours post intravenous infusion), Day 2, 3, 4/5, 8, 15, 22, 29, 43, 57, 71, 92, 120 post-infusion
Population: Pharmacokinetic analysis population included all participants who received study medication, had no protocol violations and at least one plasma tanezumab concentration.
Measure: Geometric Mean (Standard Deviation); unit: microgram/milliliter (mcg/mL)
Arm/Group | Tanezumab 10 mcg/kg | Tanezumab 25 mcg/kg | Tanezumab 50 mcg/kg | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg
Number analyzed (Participants) | 6 | 5 | 5 | 6 | 6
microgram/milliliter (mcg/mL) | 0.309 (0.0524) | 0.681 (0.2288) | 1.053 (0.1348) | 2.395 (0.3390) | 4.789 (0.6948)

57. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) - Part 1
Time Frame: as for outcome 56
Population: as for outcome 56
Measure: Median (Full Range); unit: Hour
Arm/Group | Tanezumab 10 mcg/kg | Tanezumab 25 mcg/kg | Tanezumab 50 mcg/kg | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg
Number analyzed (Participants) | 6 | 5 | 5 | 6 | 6
Hour | 0.334 [0.167 to 1.00] | 0.500 [0.167 to 24.0] | 1.00 [0.183 to 4.03] | 0.750 [0.167 to 1.00] | 0.750 [0.217 to 12.0]

58. Secondary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0-infinity)] - Part 1
Description: AUC (0-infinity) is defined as the area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-infinity). It is obtained from AUC (0-t) plus AUC (t-infinity).
Time Frame: as for outcome 56
Population: Pharmacokinetic analysis population included all participants who received study medication, had no protocol violations and at least one plasma tanezumab concentration. Here, 'overall number of participants analyzed' signifies those who were evaluable for this measure.
Measure: Geometric Mean (Standard Deviation); unit: microgram*hour/milliliter (mcg*hr/mL)
Arm/Group | Tanezumab 10 mcg/kg | Tanezumab 25 mcg/kg | Tanezumab 50 mcg/kg | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg
Number analyzed (Participants) | 6 | 4 | 5 | 5 | 6
microgram*hour/milliliter (mcg*hr/mL) | 72.05 (36.317) | 157.5 (25.586) | 312.4 (38.837) | 851.8 (281.61) | 1885 (377.43)

59. Secondary Outcome: Area Under The Curve From Time Zero to Last Quantifiable Concentration (AUClast) - Part 1
Description: AUClast is defined as the area under the plasma concentration time-curve from zero to the last measured concentration.
Time Frame: as for outcome 56
Population: as for outcome 56
Measure: Geometric Mean (Standard Deviation); unit: mcg*hr/mL
Arm/Group | Tanezumab 10 mcg/kg | Tanezumab 25 mcg/kg | Tanezumab 50 mcg/kg | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg
Number analyzed (Participants) | 6 | 5 | 5 | 6 | 6
mcg*hr/mL | 63.19 (32.747) | 183.8 (155.82) | 303.5 (37.119) | 855.5 (247.71) | 1825 (319.30)

60. Secondary Outcome: Volume of Distribution (Vz) - Part 1
Description: Vz is defined as the the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug.
Time Frame: as for outcome 56
Population: as for outcome 58
Measure: Geometric Mean (Standard Deviation); unit: milliliter per kilogram (mL/kg)
Arm/Group | Tanezumab 10 mcg/kg | Tanezumab 25 mcg/kg | Tanezumab 50 mcg/kg | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg
Number analyzed (Participants) | 6 | 4 | 5 | 5 | 6
milliliter per kilogram (mL/kg) | 51.10 (16.636) | 67.52 (30.705) | 71.08 (10.874) | 60.21 (8.9428) | 84.30 (12.885)

61. Secondary Outcome: Volume of Distribution At Steady State (Vss) - Part 1
Description: Vss is defined as the the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. It is the apparent volume of distribution at steady-state.
Time Frame: as for outcome 56
Population: as for outcome 58
Measure: Geometric Mean (Standard Deviation); unit: mL/kg
Arm/Group | Tanezumab 10 mcg/kg | Tanezumab 25 mcg/kg | Tanezumab 50 mcg/kg | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg
Number analyzed (Participants) | 6 | 4 | 5 | 5 | 6
mL/kg | 49.98 (15.192) | 66.98 (23.556) | 75.56 (16.329) | 62.74 (5.6509) | 82.56 (10.740)

62. Secondary Outcome: Systemic Clearance (CL) - Part 1
Description: CL is a quantitative measure of the rate at which a drug substance is removed from the body.
Time Frame: as for outcome 56
Population: as for outcome 58
Measure: Geometric Mean (Standard Deviation); unit: milliliter/day/kilogram (mL/day/kg)
Arm/Group | Tanezumab 10 mcg/kg | Tanezumab 25 mcg/kg | Tanezumab 50 mcg/kg | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg
Number analyzed (Participants) | 6 | 4 | 5 | 5 | 6
milliliter/day/kilogram (mL/day/kg) | 3.330 (2.2806) | 3.807 (0.5984) | 3.838 (0.5086) | 2.817 (1.3324) | 2.547 (0.4058)

63. Secondary Outcome: Mean Residence Time (MRT) - Part 1
Description: MRT was calculated as area under the moment curve/area under the concentration effect curve.
Time Frame: as for outcome 56
Population: as for outcome 58
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Tanezumab 10 mcg/kg | Tanezumab 25 mcg/kg | Tanezumab 50 mcg/kg | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg
Number analyzed (Participants) | 6 | 4 | 5 | 5 | 6
days | 17.47 (8.9511) | 18.08 (4.6284) | 19.92 (3.6745) | 23.22 (6.3625) | 33.02 (6.7913)

64. Secondary Outcome: Plasma Decay Half-Life (t1/2) - Part 1
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: as for outcome 56
Population: as for outcome 58
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Tanezumab 10 mcg/kg | Tanezumab 25 mcg/kg | Tanezumab 50 mcg/kg | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg
Number analyzed (Participants) | 6 | 4 | 5 | 5 | 6
days | 12.47 (6.4305) | 12.83 (4.2500) | 12.96 (2.0194) | 15.55 (4.5725) | 23.48 (5.4138)

65. Secondary Outcome: Percentage of Participants With Positive Anti-tanezumab Antibody Test Results
Description: Human serum anti-drug antibody (ADA) samples were analyzed for the presence or absence of anti-tanezumab antibodies by using the semi-quantitative enzyme-linked immunosorbent assay (ELISA).
Time Frame: Baseline up to Day 120
Population: FAS included all participants who had received full single intravenous dose of study medication and had at least one entry of electronic diary in both pre and post treatments. It was planned to report combined data for Part 1 and 2.
Measure: Number; unit: percentage of participants
Arm/Group | Tanezumab 10 mcg/kg | Tanezumab 25 mcg/kg | Tanezumab 50 mcg/kg | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg
Number analyzed (Participants) | 15 | 15 | 15 | 16 | 6
percentage of participants | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study.
Arm/Group | Tanezumab 10 mcg/kg | Tanezumab 25 mcg/kg | Tanezumab 50 mcg/kg | Tanezumab 100 mcg/kg | Tanezumab 200 mcg/kg | Placebo
Serious Adverse Events (participants affected / at risk) | 1/15 | 1/15 | 0/15 | 0/16 | 0/6 | 0/16
Other Adverse Events (participants affected / at risk) | 8/15 | 4/15 | 9/15 | 8/16 | 6/6 | 13/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tanezumab 10 mcg/kg (N=15) | Tanezumab 25 mcg/kg (N=15) | Tanezumab 50 mcg/kg (N=15) | Tanezumab 100 mcg/kg (N=16) | Tanezumab 200 mcg/kg (N=6) | Placebo (N=16)
Atrioventricular block (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tanezumab 10 mcg/kg (N=15) | Tanezumab 25 mcg/kg (N=15) | Tanezumab 50 mcg/kg (N=15) | Tanezumab 100 mcg/kg (N=16) | Tanezumab 200 mcg/kg (N=6) | Placebo (N=16)
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Supraventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0
Ear congestion (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 1
Asthenopia (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Visual impairment (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Face oedema (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Injection site swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 2
Oedema peripheral (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Arthritis infective (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0 | 2 | 2 | 0 | 5
Trichophytosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 1
Skeletal injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 1 | 1 | 0 | 0
Blood pressure decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Blood pressure increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Electrocardiogram T wave abnormal (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Electrocardiogram T wave amplitude decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Low density lipoprotein increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
White blood cells urine positive (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Allodynia (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0
Amnesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Decreased vibratory sense (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dysaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 2 | 1 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0
Sympathicotonia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Thermohypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Haemorrhage (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.